

Protocol number: TCH-003 

A Randomized, Double Blinded, Sham controlled Clinical Study to Evaluate the Safety and Efficacy of the Nerivio Migra 1, a Neuromodulation Device, for the acute treatment of Migraine

# Pivotal prospective multi-center clinical trial

**Clinical Investigation Plan** 

NCT03361423

01/Nov/2017

### Confidentiality statement:

The following confidential information is the property of Theranica Bioelectronics. It may only be used when permission has been obtained from Theranica Bioelectronics in writing. It is not permitted to make reproductions of all or sections of this protocol.



PROTOCOL NUMBER:

A Randomized, Double Blinded, Sham controlled Clinical Study to Evaluate the Safety and Efficacy of the Nerivio Migra 1, a Neuromodulation Device, for the acute treatment of Migraine

Protocol number: TCH-003 

# CLINICAL CLINICAL INVESTIGATION PLAN

## **STUDY TITLE:**

# A Randomized, Double Blinded, Sham controlled Clinical Study to Evaluate the Safety and Efficacy of the Nerivio Migra 1, a Neuromodulation Device, for the acute treatment of Migraine

**TCH-003** 

| REVISION: | 1.0 | | |
|---|---|---|---|
| RELEASE DATE: | 01/Nov/20 | 017 | |
| DEVICE: | Nerivio Mi | gra 1, a Neuromodulator of migraine | device for the acute |
| PRINCIPAL INVESTIGATO | ors: TBD | | |
| Sponsor: | Theranica | Bioelectronics | |
| | 45 HaMela | akha st, Netanya, Israel | |
| CONTACT DETAILS: | Dagan Har | ris, VP Clinical & Regulato | ory |
| | Tel: +972.7 | 72.390.9758 | |
| | Fax: + 972. | 72.390.9762 | |
| | Mobile: +9 | 72-0542220121 | |
| | Емаіl: <u>dag</u> | anh@theranica.com | |
| APPROVED BY: | Position: | DATE: (DDMMYY) | SIGNATURE: |
| | | // | |
| | | , , | |
| | | //_ | |




# **Version control table**

| Rev.<br>no. | Change rationale | Date |
|-------------|-----------------------------------------------|--------------|
| 1.0 | initial version for FDA pre-submission review | Oct, 1, 2017 |



Protocol number: TCH-003 

The sponsor of this study, Theranica Bioelectronics Ltd, manufacturer of the Nerivio Migra device for the acute treatment of migraine, states the following:

- a) This study will be conducted in compliance with the protocol (after being approved by the local IRB/EC and, if required, by the relevant health care agencies), US 21 CFR Parts 50, 54, 56 and 812, 45 CFR Part 46, national laws and regulation concerning clinical trials, the Good Clinical Practices (GCP) set forth in ISO 14155 (2011) standard and the ethical principles that have their origin in the Declaration of Helsinki.
- b) The Protocol, Informed Consent Form (ICF), patient's information material, and advertising material (if applicable) will be submitted and approved by the ethics and regulatory authorities, and any request by the IRB/EC or regulatory agencies will be complied with. Approval will be obtained prior to enrollment of any patients.
- c) Adequate insurance policy will be held valid for the entire study duration as well as for the discovery period required per local regulation.
- d) The study will be registered with CLINICALTRAIL.GOV



Protocol number: TCH-003 

# **Protocol Signature Page for Principal Investigator**

The signing of this Clinical Investigation Plan (CIP) by the Principal Investigator signifies that the contents have been laid down in full agreement and that the study will be conducted per this CIP, its amendments, the clinical trial agreement and the applicable regulatory requirements.

The Principal Investigator confirms that written Institutional Review Board (IRB) Ethics Committee approval for the amended CIP will be obtained prior to commencing with data collection. This approval must be in the Principal Investigator's name and a copy sent to Theranica Bioelectronics. Additionally, the Principal Investigator must sign the declaration below:

I will provide copies of this CIP and all pertinent information to the study personnel under my supervision. I will discuss this material with them and ensure they are fully informed regarding the conduct of the Study.

| Principal Investigator's Signature | Date |
|---------------------------------------|--------|
| Principal Investigator's Printed Name | _ |
| Site Name | Site # |



Protocol number: TCH-003


# **Contents**

| 1 | | | S | |
|---|---|---|---|---|
| 2 | $\mathbf{B}_{A}$ | | OUND | |
| | 2.1 | | CTION | |
| 3 | ID | | ICATION AND DESCRIPTION OF THE DEVICE | |
| | 3.1 | | O USE | |
| | 3.2 | | CE | |
| | 3.3 | | ICATION | |
| | 3.4 | | DUTPUT | |
| | 3.5 | | TION AND VALIDATION | |
| | 3 | | erformance testing | |
| | 3 | | oftware validation | |
| | 3.6 | | E OF OPERATION | |
| | 3.7 | | ATION OF THE MEDICAL DEVICE | |
| | 3.8 | | TIONS FOR USE | |
| | 3.9 | | y of Necessary Training | |
| 4 | | | NARY INVESTIGATIONS AND JUSTIFICATION FOR THE STUDY DES | |
| | 4.1 | | S PRE-CLINICAL EXPERIENCE | |
| | 4.2 | | S CLINICAL EXPERIENCE | |
| | 4.3 | | Investigation Risks and Benefits | |
| 5 | | | VES & HYPOTHESES | |
| | 5.1 | | E | |
| | 5.2 | | SIS | |
| 6 | | | OF THIS CLINICAL STUDY | |
| | 6.1 | | TON | |
| | 6.2 | | ES TO MINIMIZE BIAS | |
| | 6.2.1 | | OMIZATION | |
| | 6.2.2 | | EDURES TO ENSURE BLINDING | |
| | 6.3 | | NDPOINTS | |
| | 6.4 | | S AND TIMING OF ASSESSING, RECORDING AND ANALYZING VARIABLES | |
| | 6.4.1 | | OF DATA | |
| | 6.4.2 | CLINIC | CAL STUDY VARIABLES AND DATA CAPTURE TOOLS | |
| | 6.4 | 4.2.1 | Start attack/episode PRO feedback data | |
| | 6.4 | 4.2.2 | 2h PRO | |
| | 6.4 | 4.2.3 | 48h PRO | |
| | 6.4.3 | | ODS AND TIMING OF ASSESSING, RECORDING AND ANALYZING VARIABLES | |
| | 6.4.4 | | FLOW AND MANAGEMENT | |
| | 6.4.5 | | EDURES FOR REVIEW OF DATA | |
| | 6.4.6 | DATA | MONITORING COMMITTEE | 46 |
| | 6.4.7 | Total | L EXPECTED DURATION OF THE CLINICAL INVESTIGATION | 47 |
| | 6.5 | SUBJECTS | | 47 |
| | 6.5.1 | INCLU | SION CRITERIA | 47 |
| | 6.5.2 | Exclu | JSION CRITERIA | 47 |
| | 6.5.3 | CONT | RAINDICATIONS | 48 |
| | 6.5.4 | Nume | BER OF SUBJECTS | 48 |
| | 6.5.5 | EXPEC | TED STUDY DURATION FOR EACH SUBJECT | 48 |
| | 6.5.6 | POINT | r of Enrollment | 48 |
| | 6.5.7 | PATIE | NT WITHDRAWAL CRITERIA | 48 |
| | 6.5.8 | HAND | DLING OF WITHDRAWALS | 49 |



Protocol number: TCH-003 

| | 6.5.9 | PATIENT LOST TO FOLLOW-UP | 49 |
|---|---|---|---|
| | 6.5.10 | ENROLLMENT PERIOD | 49 |
| | 6.5.11 | PROCEDURES FOR REPLACEMENT OF SUBJECTS | 49 |
| | 6.6 S | TUDY RELATED PROCEDURES | 50 |
| | 6.6.1 | GENERAL | 50 |
| | 6.6.2 | VISIT AND ASSESSMENT SCHEDULE | 50 |
| | 6.6.3 | ACTIVITIES PERFORMED BY SPONSOR REPRESENTATIVES. | |
| | 6.7 N | MONITORING PLAN | |
| 7 | | TISTICAL CONSIDERATIONS | |
| | 7.1 S | TUDY DESIGN AND AIM | 52 |
| | 7.2 S | TUDY VARIABLES | 52 |
| | 7.2.1 | PRIMARY PERFORMANCE VARIABLE | 52 |
| | 7.2.2 | SECONDARY PERFORMANCE VARIABLES | 52 |
| | 7.2.3 | EXPLORATORY PERFORMANCE VARIABLES | 52 |
| | 7.2.4 | SAFETY VARIABLES | 52 |
| | 7.3 S | TUDY HYPOTHESIS | 52 |
| | | AMPLE SIZE ESTIMATION | |
| | | PEFINITION OF ELIGIBLE TREATMENT | |
| | 7.6 In | NTERIM ANALYSIS | 53 |
| | | ANDOMIZATION | |
| | | NALYSIS SETS | |
| | | TATISTICAL ANALYSES – (TBD) | |
| | 7.9.1 | GENERAL CONSIDERATIONS | |
| | 7.9.2 | SIGNIFICANCE LEVELS AND HANDLING OF TYPE I ERROR | |
| | 7.9.2.1 | | |
| | 7.9.2.2 | | |
| | 7.9.3 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| | 7.9.4 | DISPOSITION OF PATIENTS. | |
| | 7.9.5 | PERFORMANCE ANALYSES | |
| | 7.9.6 | SAFETY ANALYSIS: | |
| | 7.9.7 | HANDLING OF MISSING DATA | |
| | 7.10 | Pooling | |
| 8 | _ | ΓA MANAGEMENT | |
| | | NATA CAPTURE | |
| | 8.1.1 | | |
| | | PATA QUALITY ASSURANCE | |
| | | LECTRONIC SIGNATURES. | |
| | | ERIFICATION, VALIDATION AND SECURING OF ELECTRONIC DATA CAPTURE SYSTEM | |
| | | ECORDS AND DATA RETENTION | |
| | | OTHER ASPECTS OF CLINICAL QUALITY ASSURANCE | |
| 9 | | ENDMENTS TO THE CLINICAL INVESTIGATION PLAN | |
| ,<br>10 | | NICAL INVESTIGATION PLAN DEVIATIONS | |
| 10 | 10.1 | PROCEDURES FOR RECORDING, REPORTING AND ANALYZING PROTOCOL DEVIATIONS | |
| | 10.2 | NOTIFICATION REQUIREMENT AND TIMELINES | |
| 11 | - | VICE ACCOUNTABILITY | |
| 12 | | TEMENTS OF COMPLIANCE | |
| 13 | | ORMED CONSENT PROCESS | |
| 14 | | VERSE EVENTS | |
| | 1/11 | CHARACTERISTICS OF AN ADVERSE SVENT | 66 |




| 14.1 | 1.1 Severity of the Adverse Event | 66 |
|---|---|---|
| 14.1 | 2 Relationship of an AE and SAE to the Study Device | 66 |
| 14.2 | DEFINITIONS OF ADVERSE EVENT AND ADVERSE DEVICE EFFECT | |
| 14.3 | DEFINITION OF SERIOUS ADVERSE EVENT | 67 |
| 14.4 | DEVICE DEFICIENCY | 67 |
| 14.5 | TIME-FRAME FOR INVESTIGATOR REPORTING AE TO SPONSOR, EC, RA | 67 |
| 14.6 | ADVERSE EVENT REPORTING FORMS | 68 |
| 14.7 | FORESEEABLE COMPLICATIONS AND ANTICIPATED ADVERSE DEVICE RELATED EFFECTS | 68 |
| 14.8 | SAFETY MONITORING AND ADJUDICATION OF ADVERSE EVENTS | 69 |
| 15 VU | LNERABLE POPULATION | 70 |
| 16 EA | RLY TERMINATION OF THE CLINICAL INVESTIGATION | 71 |
| 16.1 | CRITERIA AND ARRANGEMENTS | 71 |
| 16.2 | REQUIREMENTS FOR PATIENT FOLLOW-UP IN CASE OF WITHDRAWAL | |
| 17 PUI | BLICATION POLICY | 72 |
| | FIENT CONFIDENTIALITY & DATA PROTECTION | |
| | IDELINES AND APPLICABLE DOCUMENTS | |
| | FERENCES | |
| | RONYM LIST | |
| | IX A. STIMULATION PROGRAMS | |
| <b>APPEND</b> | IX B. CASE REPORT FORMS LIST AND DRAFT CRF QUESTONS | 80 |



Protocol number: TCH-003 

# 1 SYNOPSIS

| Title | A Randomized, Double Blinded, Sham controlled Clinical Study to Evaluate the Safety and Efficacy of the Nerivio Migra 1, a Neuromodulation Device, for the acute treatment of Migraine |
|---|---|
| Sponsor | Theranica Bioelectronics Ltd. 45 HaMelakha st, Netanya, Israel |
| Investigational<br>Device | Nerivio Migra, a neurostimulation device, is intended for the acute treatment of migraine with or without aura in patients 18 years of age or older. The device delivers transcutaneous electrical stimulation below pain threshold to the patient's upper arm. The level of generated stimuli is similar to other FDA approved electro- stimulation devices. The treatment is self-administered and controlled by a dedicated smartphone application. It is believed to alleviate pain through conditioned pain modulation. |
| Study Design | A prospective, randomized (1:1), double-blind, sham-controlled trial. The study will be conducted in three stages; two mandatory stages, and one optional stage. Stage One - Roll-in: Eligible participants will be trained to use a smartphone migraine diary application. After the enrollment visit, participants who successfully completed training will report all their migraine attacks using the smartphone application for up to one month. Only patients who properly report at least 2 and no more than 8 migraine attacks, with a compliance rate as defined in section 6.1, will continue to the next stage. Stage Two - Parallel arm, double-blind treatment stage: Participants who meet the entry requirements will be randomized to an active Nerivio Migra or an identically looking sham device. They will be trained to use the device for treatment and provide feedback via the smartphone application. The active/sham ratio is 1:1. Following successful completion of training, subjects will be asked, to apply the device and administer treatment for every migraine attack they experience, at the onset of their migraine attack. Subjects will be asked to report the results of every treatment, using the smartphone application, at the times preset in the application. Subjects will be asked to carry the device and their smartphones with them at |
| | all times, and to make a reasonable effort to keep their smartphone charged and connected to the Internet at all times. |




| | The first treated attack in the double-blind treatment stage is considered a "run-in test" treatment; its purpose is to verify compliance. This "run-in test" is only included in the safety endpoint analysis. It will not be included in the primary and secondary performance endpoints analysis. |
|---|---|
| | Stage Two will end after four (separate) treated migraine attacks, (excluding the "run-in test" attack), or one month (whichever is achieved first). |
| | Stage Three (optional, by subject request only) - Open label extended |
| | treatment: |
| | Following the completion of double-blind stage of the study, all subjects will be offered a 2-month open label period using the active device. |
| Objectives | To demonstrate the safety and effectiveness of the Nerivio Migra electro stimulation device for the reduction of migraine headache during an attack of migraine with or without aura. |
| Safety Endpoints | Adverse events related or unrelated to the study device. |
| | 2. Treatment tolerability |
| Primary | Reduction of migraine headache: |
| Performance | The proportion (%) of patients reporting reduction in their pain level 2 hours post- |
| Endpoint | treatment without rescue medications from severe or moderate to mild or no |
| | pain, or from mild to no pain, in their first treated migraine attack (excluding the "run-in test" treatment). |
| Secondary | · |
| Performance | 1. MBS Relief: Proportion (%) of patients reporting, 2 hours post-treatment, freedom from |
| | their most bothersome migraine-associated symptom (MBS) other than a |
| Endpoints | headache, in their first treated migraine attack (excluding the "run-in test" |
| | treatment). MBS may be nausea, photophobia, phonophobia or allodynia – |
| | as defined by each subject at the beginning of the treatment. |
| | Reduced Migraine Headache AND MBS Relief: |
| | Proportion (%) of patients reporting, 2 hours post treatment response to |
| | both the primary and the first secondary endpoints. |
| | 3. Pain-free at 2 hours: The proportion (%) of subjects reporting freedom from migraine pain at 2 hours post-treatment without medications in their first treated migraine attack (excluding the "run-in test" treatment). |



Protocol number: TCH-003 

| Exploratory |
|-------------|
| Performance |
| Endpoints |

- 1. Sustained pain-free 48 hours with **single** use of the device:
  The proportion (%) of subjects reporting pain-free at 2 hours, and no return of any pain or use of rescue/acute medication, or reuse of device between 2 hours and 48 hours, in their first treated migraine attack (excluding the "run-in test" treatment).
- 2. Sustained Headache Reduction for 48 hours with single use of the device: The proportion (%) of subjects reporting treatment response 2 hours post-treatment without rescue medications, and no return to baseline level of pain at time of treatment, or use of rescue/acute medication, or reuse of device between 2 hours and 48 hours, in their first treated migraine attack (excluding the "run-in test" treatment).

Treatment response is defined as:

- pain level reduction from moderate or severe at baseline to mild or none, OR:
- o pain level reduction from mild to no pain.
- 3. Sustained pain-free 48 hours with **reuse** of device
  The proportion (%) of subjects reporting pain-free at 2 hours, and no
  return of any pain or use of rescue/acute medication except for reuse of
  device between 2 hours and 48 hours, in their first treated migraine attack
  (excluding the "run-in test" treatment).
- 4. Sustained Headache Relief 48 hours with **reuse** of the device:
  The proportion (%) of subjects reporting Treatment Response at 2 hours, and no return to baseline level of pain at time of treatment, or use of rescue/acute medication except for reuse of device between 2 hours and 48 hours, in their first treated migraine attack (excluding the "run-in test" treatment).

Treatment response is defined as:

- pain level reduction from moderate or severe at baseline to mild or none, OR:
- o pain level reduction from mild to no pain.
- 5. Sustained relief of MBS with a **single** use of the device
  The proportion (%) of subjects reporting freedom from MBS at 2 hours,
  and no return of MBS, or use of rescue/acute medication between 2 hours
  and 48 hours, in their first treated migraine attack (excluding the "run-in test" treatment).



| Protocol number: TCH-003 | age <b>12</b> of <b>94</b> |
|--------------------------|----------------------------|
|--------------------------|----------------------------|

| , |
|---|
| <ol> <li>Sustained relief of the MBS with reuse of the device: Proportion (%) of patients reporting, 48 hours post the first treatment, freedom from their most bothersome migraine-associated symptom other than headache (MBS), possibly with reuse of the device, in their first treated migraine attack (excluding the "run-in test" treatment). </li> <li>Within-patient consistency of the primary endpoint in subsequent treatments: The repeatability of migraine headache reduction, as described in the primary endpoint definition, in subsequent treated attacks. Thus, this endpoint measures the % of patient responding to the primary endpoint in at least 50% of their treated attacks (excluding the run-in </li> </ol> |
| attack |
| Adults 18-75 years old meeting International Headache Society criteria (ICDH3) for migraine with and without aura, who are reporting 2-8 migraine attacks per month. |
| up to 270 patients with evaluable data, equally distributed between US and non-US sites |
| 1. Subjects age 18-75 years old. |
| 2. Subjects meet the ICHD-3 diagnostic criteria for migraine with or without aura |
| 3. Subjects report 2-8 migraine attacks per month. |
| 4. Stable migraine preventive medications in the last two months prior to recruitment (No change in usage or dosage). |
| 5. Subjects must be able and willing to comply with the protocol |
| 6. Subjects must be able and willing to provide written informed consent |
| <ol> <li>Subject has other significant pain, medical or psychologic problems that in the opinion of the investigator may confound the study assessments</li> <li>Subject has an implanted electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagus nerve neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator cochlear implant, Sphenopalatine ganglion stimulator or Occipital nerve stimulator).</li> </ol> |
| 3. Subject has known uncontrolled epilepsy. |
| 4. Any use of Cannabis including medical use. |
| 5. Subject has >10 headache days per month. |




- 6. Subject has undergone nerve block (occipital or other) in the head or neck within the last 2 weeks.
- 7. Subject is participating in any other clinical study.
- 8. The subject does not have the basic cognitive and motor skills needed to operate a smartphone.
- 9. Pregnant, or trying to get pregnant
- 10. Subject is experiencing a menstrually related migraine
- 11. Received OnabotulinumtoxinA or any botulinum toxin injections for migraine within the previous month
- 12. Received parenteral infusions for migraine within the previous 2 weeks.
- 13. Subject participated in a previous study with the Nerivio Migra 1 device

<u>Note</u> - Females of child bearing potential must have a negative pregnancy test and must be willing to use adequate contraception during the study

### **Study Procedures**

### **Enrollment visit:**

Following successful eligibility screening, enrollment interview and signing of informed consent, participants will be trained in the Nerivio Migra software application in its "diary" mode. The application will be installed on their smartphones (or smartphones provided by the clinic, if the patient does not have a compatible smartphone).

Subjects will complete a baseline questionnaire including the frequency and severity of migraine attacks, usual most bothersome symptom, usage of preventive and acute medications and devices.

#### Roll-in stage:

After the enrollment visit, patients will be asked to report each and every migraine attack with the application. (These reports will be collected).

Participants who successfully complete the roll-in stage with at least 2 but no more than 8 migraine attacks, with complete and prompt reporting and compliance rates as defined in section 6.1, will be eligible for randomization.

### Randomization visit:

Patients will be randomized and provided with an active Nerivio Migra or an identically looking sham device. Then they will be trained to use the device and provide feedback via the smartphone application.



Protocol number: TCH-003 

### Treatment stage:

After the randomization visit, patients will be asked to treat all their migraine attacks with the device, if, and only if, they can apply the device immediately after the onset of the migraine attack symptoms and no later than 60 min, and report through the application, at the preset times on the application. Patients will be asked to keep the device and their smartphone with them at all times and make a reasonable effort to keep the smartphone charged and connected to the Internet.

Patients will be asked not to use rescue medications during the first two hours after the start of treatment. Taking rescue medication in this time period is considered a major protocol violation. Patients will record their medication use in the smartphone application.

At the beginning of treatment, two, and 48 hours later, each participant will be prompted by the application to rate their migraine pain level using Pain Grades Scale with values 0-3 (no pain, mild, moderate, severe), and other symptoms of the migraine attack: aura, nausea, photophobia, phonophobia and allodynia.

In case of failure to provide feedback regarding pain level posttreatment, alerts will be generated by the Electronic Data Collection system, and telephone follow-up inquiries will be performed by study investigator staff.

Two hours after treatment and completing the post two-hour feedback, subjects will be able re-treat the attack – if they choose so - by re-using the Nerivio Migra device as often as they want.

After completing up to 4 qualified treatment, or 1 month from the randomization visit (whichever happens first) subjects will stop using their device until their next visit.

### Open Label visit:

Subjects will fill an end of study questionnaire, which includes patient global impression of the change in their migraine experience with the device, blinding questionnaire, and usability assessment.

After completing the questionnaire, subjects will be offered an active which they will be able to use for the next two months.




| | Onen Lahel extension: |
|---|---|
| | Open Label extension: All treatments will be recorded and monitored (identical to the dual-arm |
| | treatment phase). Adverse events will also be recorded. |
| | Final visit: (This can occur at the open label visit if patients do not want to |
| | continue to use the device): |
| | At the end of the Open-Label extension, patients will return the device to the clinic. |
| | Adverse events will be collected throughout the study. |
| Study Duration | Duration for each patient will be approximately two months – up to one |
| | month of roll-in stage and up to one month or treatment of up to four |
| | qualified migraine attacks (whichever is achieved first). |
| | An optional open-label extension of two months is available. |
| Qualified | Qualified treatments must meet ALL the following criteria: |
| Treatments | The patient had at least 48 consecutive hours without migraine |
| | headache prior to treatment. |
| | 2. Treatment is started no later than 60 minutes post the onset of |
| | migraine symptoms. |
| | 3. Treatment lasted at least 30 (continuous) minutes. |
| | 4. No pain medications were used from 24 hours prior the onset of |
| | the migraine, until 2 hours after the start of the treatment. |
| | 5. The patient completed and reported the post 2-hour treatment |
| | questionnaire through the application. |
| Major Protocol | The following will be considered major protocol violations: |
| Violations | Taking rescue medication within the two hours of starting |
| | treatment. Such treatments will be considered non-qualified. |
| | 2. Starting the treatment more than 60 mins after the onset of |
| | migraine symptoms. Such treatments will be considered non- |
| | qualified. |
| | 3. Not completing 30 minutes of treatment. Such treatments will be |
| | considered non-qualified. |
| Sample Size | Up to 270 subjects will be recruited to this study |
| Data Analysis | Data management function will be supported by a cloud-based EDC system |
| | (Clear Clinica, Modi'in, Israel). Clear Clinica provides services for collection |
| L | l |



Protocol number: TCH-003


and remote monitoring of clinical trials data, compliant with HIPAA and 21 CFR Part 11.

EDC portals with secure authorized access will be made available to the site personnel, as well as to the study monitor.

Data captured by clinical personnel will be entered directly into prespecified eCRF screens by site personnel. Data from paper sources will be entered into the study database. Automatic data checks will be implemented for the majority of entry fields to provide an opportunity for resolving data inconsistencies as close as possible to real time.

Data collected onto the smartphone application will be directed to a secure cloud-based database where it will undergo analysis aimed at detection of missing data and other inconsistencies.

Activities such as repeatedly aborted programs, missing feedbacks, inconsistent stimulation intensity adjustments, and similar, will be communicated to research coordinator of the corresponding site, using participants' ID codes. Missing data will be identified automatically, and queries will be generated to participants and corresponding site study coordinator.

### Statistical analysis

### **Analysis Sets**

1. Intent to Treat analysis set (ITT)

The ITT analysis set includes all patients who are randomized and treat at least one attack.

2. Modified Intend to Treat analysis set (mITT)

The mITT analysis set includes all patients who are randomized and treat at least one attack (excluding the" run-in test" attack) within 1 hour from the attack onset.

3. Per-Protocol analysis set (PP)

The PP analysis set includes patients who are randomized and treat at least one attack (excluding the "run-in test" attack), which conforms with the protocol instructions:

- Treatment starts within one hour from attack onset.
- No rescue medication (or pain medication) is consumed within the 2 hours after start of treatment.
- The treatment is not aborted prematurely (i.e., before the first 30 minutes).
- No Pain medication 24h prior migraine onset



Protocol number: TCH-003 

Statistical Analysis of Analysis Sets

The ITT analysis set will serve as the main set for safety assessments.

The mITT analysis set for all performance assessments.

The primary and secondary performance assessments will also be performed on the PP analysis set as a sensitivity analysis.




### 2 BACKGROUND

### 2.1 Introduction

Migraine is a common neurologic with attacks of headache and associated symptoms such as nausea, vomiting, phono and photophobia. Migraine can lead to substantial functional impairment [1]. The recent Global Burden of Disease Study 2010 (GBD2010), conducted by the World Health Organization, estimates a worldwide prevalence of migraine of 14.7%, ranking it third place among the most common diseases and at the seventh place among specific causes of disability and top of all neurological disorders as cause of total years lived with disability [1]. The pathophysiology of migraine is becoming understood [2]. Current approach to migraine treatment is predominantly pharmacological [3].

Transcutaneous electrical stimulation (ES) is a non-invasive technique that delivers series of weak electrical pulses to patient's skin. ES has been used for decades for treatment of many painful conditions [3, 4]. In general, the stimulation is applied adjacent to, or at least within the dermatome of the painful body site. Recent evidence suggests that electro stimulation is effective in providing relief for chronic headaches including migraine. It is tolerable by patients and associated with no adverse effects [4-6]. There are currently two approved non-invasive devices intended for providing migraine relief via transcutaneous electro stimulation. The first device, Cefaly, is used for acute and preventive treatment migraines, was developed by STX-Med [4]. The device applies electro stimulation to the forehead, within the trigeminal nerve territory. The second device, GammaCore, developed by ElectroCore [6], vagus nerve stimulation is approved for marketing in Europe and is used for treatment of migraine pain. It is approved in the US for the acute treatment of episodic cluster headache. Both devices deliver stimulation at relatively low intensity (16mA). Both devices target electro stimulation to major specific nerves in close proximity to patient's head. Both trigeminal and vagus nerves are responsible for multiple functions of major importance. The list includes, but is not limited to, facial sensation, biting, chewing for trigeminal nerve; heart rate, sweating and speech for vagus nerve.

These commercially available treatment approaches are associated with some usability challenges (Cefaly device is mounted on forehead and the GammaCore is hand held throughout the treatment session but only 90 seconds).

There exists a need for additional non-pharmacological solutions for migraine treatment.



Protocol number: TCH-003 

### 3 IDENTIFICATION AND DESCRIPTION OF THE DEVICE

Theranica has developed Nerivio Migra ("Migra" or "the device"). Nerivio Migra is intended for the acute treatment of migraine with or without aura in patients 18 years of age or older. It is self-applied to the upper arm. Treatments are self-administered by the user at the onset of a migraine attack. The device delivers extra cephalic transcutaneous electrical stimulation below the pain threshold to the skin of the upper arm at the onset of a migraine attack. Nerivio Migra is operated via a mobile application.

Nerivio Migra utilizes electro stimulation to achieve conditioned pain modulation (CPM). Conditioned Pain Modulation (CPM) [7] is a paradigm used in pain research, in which a "conditioning" (also referred to as secondary) stimulus is applied to influence the subject's perception of a "conditioned" (primary) painful stimulus, delivered (or originating) at a different y location. Based on diffused noxious inhibitory control (DNIC) mechanism [14], and sometimes referred to as "pain inhibits pain" principle, CPM evokes an endogenous analgesic mechanism. The modulatory effect is over the whole body, and can be induced anywhere in the body. This approach allows applying the conditioning stimuli away from the painful site.

The conditioning stimulus is given at an intensity which is well felt, but below the pain threshold. Experimental human data shows that in the majority of tested subjects, a conditioning stimulus which is slightly lower than pain threshold is sufficient to activate CPM [8, 9]. This is probably due to different summation requirements of the brainstem pain modulation centers and of the cortex; more intensive peripheral nociceptive activity is needed for the cortex than for the brainstem. The 'inhibitory power' activated by CPM via this peripheral non-painful stimulation is limited. It is most effective when used migraine headache onset, when activity of the nociceptive pathways is still just starting, and may be related to lack of central sensitization. Central sensitization often develops during the first two hours of the migraine attack; this explains the benefit of early treatment. [10] Thus, treatment early in the attack is expected to be more effective.

The device delivers electrical currents that are within the range of FDA approved battery operated Transcutaneous electrical nerve stimulation (TENS) devices to treat pain [18, 19].

The use of TENS has proved effective in clinical studies and its safety is well established [15-17]. Multiple TENS devices are being marketed for over-the-counter use for a wide range of indications and anatomical locations. Many approved devices are used to treat chronic conditions.

Two main groups of electro stimulation protocols have been described and evaluated for pain relief: high frequency (80-200Hz) and low frequency (1-5Hz) [18]. Nerivio Migra operates in high frequency domain.

To the best of our knowledge this is the first device based on application of electrical stimulation to treat migraine headache through conditioned pain modulation allowing for the application of the stimulator remotely to head and neck.

The device is comprised of 3 main components: (1) Arm-band with attached electrodes, (2) Electronics case and (3) Software including Firmware and Mobile Application software to be run on a mobile platform. Each of these components is briefly described below.



Protocol number: TCH-003


### 3.1 Intended Use

The Nerivio Migra device is intended for the acute treatment of migraine with or without aura in patients 18 years of age or older.

The Nerivio Migra is indicated to be applied within no more than 60 minutes from migraine symptoms onset. The Nerivio Migra is indicated for self-administration in home setting.

### 3.2 The Device

The Device is a fully integrated unit similar in appearance to an armband. The device includes an arm band, electronic circuitry and battery contained in a plastic case, and a pair of electrodes with hydrogel (**Figure 1**).



Figure 1. - Internal side of Nerivio Migra device

The armband is based on biocompatible materials and comply with the biocompatibility requirements (according to ISO 10993 part 1- biological evaluation for medical devices). It is thin and stretchable, as to not impede the user's movement. The Velcro strip allows convenient placement of the device at intended arm area for variety of arm sizes.

A pair of electrodes is attached to the internal side of the armband. The 5cm x 5cm Ultra Slim Electrodes with multistick gel (Model SN2020) are manufactured by Axelgaard Manufacturing Co. Ltd (Fallbrook CA, USA). The electrodes are incorporated into the armband and are not to be replaced by participants throughout the course of the study.



Protocol number: TCH-003 

The plastic case, made of non-flammable ABS type plastic, is placed on the armband in a manner that does not result in its contact with the body. The plastic case contains the device's electronics circuitry. It is attached to the external surface of the armband and wired to the electrodes that are housed on the inside of the armband. The case dimensions are 10cm x 5cm x 1.5cm.

The electronic circuitry housed within the plastic case contains a small printed circuit board (PCB) with the electronics components that are needed to generate and operate the electro stimulation functions (delivered via the electrodes) as well as the wireless communication with the user's smartphone or tablet (via standard Bluetooth protocol). The PCB connects to a battery located inside the case, and is wired to the pair of stimulation electrodes.

The outer part of the case contains an on/off switch and LED indicator of working mode (**Figure 2**).



Figure 2. - External side of Nerivio Migra device

The device includes current source circuitry that ensures steady stimulation current output. The current output is limited by the current source hardware design to 60mA. The output voltage is further limited by the power supply hardware design to 60V.

The device uses a controlled current source to output steady and controlled current via a pair of electrodes. The stimulation program is stored in device memory. The waveform is generated by the Pulse Generator unit and controlled by a programmable microcontroller ( $\mu$ CPU) to follow preset stimulation program parameters. Intensity of the output current can be controlled via mobile app software by Bluetooth wireless connection (BT/BLE). Once stimulation has been started by user, the device can operate in a stand-alone fashion without wireless connection to the mobile app software and will automatically cease stimulation after reaching the program's time limit.

The provided battery is sufficient to provide power required for stimulation throughout the duration of the whole experiment. The device will not be connected to power outlet by study participants.

An ID sticker used to uniquely identify the device, as well as assist with a quick Bluetooth pairing is placed on the external side of the device.



Protocol number: TCH-003


# 3.3 The Application

Activation, control over stimulation intensity and termination of stimulation are performed via a dedicated smartphone application developed by Theranica and installed on the user's cell phone.

The Nerivio Migra Application provides user interface for operating and managing the device, means for collecting Patient Reported Outcomes (PRO) and the link to the secure cloud and study database (DB). Captures of main Application screens are shown in **figure 3**.

The Application is installed from a standalone APK file, fully independent and distributable; implementation for Android only (4.1 and above).

- Upon activation, the Application shows the main window with the following options for the user to select:
  - Connection handles the Bluetooth connection to the device
  - Diary/Treatment collects information regarding migraine symptoms, controls the stimulation programs, as well as user feedback regarding the treatment
  - Help provides online help to the user
  - Switch to treatment register the patient and the device for the treatment stage
- The Application logs and records every operation of the device into NVM on the Smartphone. Subsequently, this information is also relayed to the Cloud (see **Figure 7**).
- The Application is able to query device battery status and notify the user of its condition.
- Supports menus and display language in Hebrew and English (according to phone's language set)
- Supports PRO collection
- Keeps logs of the actions performed by the user, including:
  - Device's connection and disconnection
  - Activation and deactivation periods
  - User stimulation intensity adjustments
  - Feedback from the user (before, during and after activation)









Figure 3. - Application screens. Left to right: start screen, main menu, connectivity screen, treatment management screen



Protocol number: TCH-003 

# 3.4 Energy output

Output parameters of the Migra are similar to those of other TENS devices previously cleared by the FDA and currently marketed for variety of indications for over the counter use.

The Nerivio Migra output parameters and its comparison to other approved devices are described in **table 1** 

| Parameter | Nerivio Migra 1 | Cefaly | Sys*Stim TENS |
|---|---|---|---|
| Mode or Program name | TENS | TENS | TENS |
| Waveform | Biphasic,<br>symmetrical | Biphasic,<br>symmetrical | Asymmetrical biphasic with zero net DC |
| Shape | Rectangular | Rectangular | Rectangular |
| Maximum output voltage (V) | | | |
| 500Ω | 30 | 8 | 92 ±20% |
| 2ΚΩ | 60 | 32 | 144 ±20% |
| 10ΚΩ | 60 | 60 | 166 ±20% |
| Maximum output current (mA) | | | |
| 500Ω | 60 | 16 | 184 ±20% |
| 2ΚΩ | 30 | 16 | 72 ±20% |
| 10ΚΩ | 6 | 6 | 17 ±20% |
| Duration of primary (depolarizing) phase (μsec) | 200 | 250 | 200μs ±10% |
| Frequency (Hz) | 100-120 | 60 | 1-80Hz ±10% |
| Maximum average power density (mW/cm²)500Ω | 3.17 | 0.017 | 12 |
| Maximum phase charge (μC) | | | |
| 500Ω | 12 | 4 | 33.5u ±10% |



| Protocol number: TCH-003 | Page <b>24</b> of <b>94</b> |
|--------------------------|-----------------------------|
|--------------------------|-----------------------------|

| Maximum current density (mA/cm², r.m.s) | | |
|-----------------------------------------|------|------|
| 500Ω | 0.50 | 2.37 |

Table 1 - Key output parameters comparison

User has control over stimulation intensity within the specified limits. A dedicated mechanism controls speed of intensity adjustment in order to protect the user from unexpectedly strong stimulation intensity variations.

# 3.5 Verification and validation

The design of the Nerivio Migra device has been verified and validated as per the design control requirements (FDA 21 CFR part 820.30 and ISO 13485). The device successfully passed basic safety and EMC tests per applicable standards (leakage current, power consumption and radiation emission) at Hermon Laboratories.

# 3.5.1 Performance testing

All features and output specifications identified in Table 1 were verified under various loading conditions meant to simulate those the device could encounter during use.

Bench tests of the device included:

- Verification of stimulation programs pulses characteristics, program duration, and stimulation intensity. The tests were performed using e\*Scope TDS3012B manufactured by Tektronix (USA).
- Mechanical testing
- Bluetooth connectivity distance and robustness
- Battery lifetime for active and passive states.

### 3.5.2 Software validation

Validation of software (smartphone application) relating to the function of the device was performed for variety of use cases providing coverage of device requirements.

#### It includes:

- Application in general
- Authorization
- Connectivity with the device
- Help / troubleshooting messages
- Programs execution



Protocol number: TCH-003 

- Activation
- Amplitude control
- User feedback
- Battery measurement
- Android version
- Logs
- Application dialogs
- Client/server communication
- Notifications
- User feedback –additional data
- Notification to switch down device

# 3.6 Principle of Operation

Once Migra is placed on the patient's arm (see **Figure 4**) at the onset of a migraine attack, the user turns the device ON and activates therapy via the Mobile Application.



Figure 4 - Nerivio Migra located on the upper arm

This target location is easily accessed independently by the patient without help and is discrete to maintain treatment privacy. The treatment delivered to the user is a weak electrical current to the skin via the electrodes.

The operation of Migra is controlled by mobile application software that was developed by the company. The application is installed and operated from the patient's smartphone device, and is used for the activation, termination and control (e.g. stimulation intensity control, status indications and more) of the device.

The communication between the Migra device and the Application software is performed wirelessly via standard Bluetooth protocol.

Duration of the stimulation program is pre-set to 45 minutes. At any point in time, however, the patient is able to stop treatment by one of three methods:




- Terminating the stimulation via the Mobile Application
- Turning off the device on/off switch located on the outer part of the armband
- Carefully removing the armband

For the study purposes, the Nerivio Migra delivers a single, pre-set, active stimulation program, or a sham program. Programs characteristics are given in Appendix A.

Device operation flow is presented in the figure 5.



Figure 5. - Device operation flow

At any moment during treatment, user can stop treatment by terminating the stimulation via the smartphone application, or by turning off the switch on the wearable unit, or by simply removing the armband.

# 3.7 Identification of the Medical Device

The medical device will be labeled for clinical investigation use only. The label includes the address of the legal manufacturer and all other essential information to allow full traceability of the medical device as per the regulatory labeling requirements.

# 3.8 Instructions for Use

Device Instructions for Use are available as a separate document to study personnel. Printed instructions for Use are handed to study participants along with the device. Electronic version of



Protocol number: TCH-003 

IFU is accessible from the Application at any time. A brief description of principle of operation can be found in sections 3.1- 3.4 above.

# 3.9 Summary of Necessary Training

General instructions and training in device use as peer the IFU will be provided to study participants at the participating sites. No specific skills are required from study participants beyond basic level of experience with general purpose Android applications. Training will be delivered by designated study personnel and will be recorded in a corresponding CRF. In addition, records of the training session will be documented in the study DB with label "training". The criteria for training effectiveness will be ability of the participant to run a training treatment session independently.

Training to the investigator and staff will be delivered by sponsor representative in a frontal session including demo and training activations. In order to provide additional support to clinical personnel, a training video clip was prepared and will be available at all training sessions for staff and participants.



Protocol number: TCH-003


# 4 PRELIMINARY INVESTIGATIONS AND JUSTIFICATION FOR THE STUDY DESIGN

### 4.1 Previous Pre-Clinical Experience

There were no animal studies with the Nerivio Migra device. Since it is applying energy output similar to that of FDA approved TENS devices, and in accordance with the application of risk management as per EN ISO14791, the necessity for such a study has been precluded. There is no valid animal model to test the effectiveness of this device.

# 4.2 Previous Clinical Experience

Sponsor has completed a prospective, randomized, double-blind, sham controlled, cross-over, multiple treatment arms single center study "Relief of migraine pain through electro stimulation" at the Neurology Department, Rambam Medical Center (Haifa, Israel). A brief summary of this pilot study protocol is provided below, along with an overview of the procedures utilized and the results observed.

### **Pilot Study Objective**

The purpose of the investigation was to evaluate the safety and performance of the Nerivio Migra for the relief of headache pain of non-chronic migraine patients with and without aura and provide comparative data regarding performance and tolerability of the evaluated treatment programs.

#### **Inclusion and Exclusion Criteria**

#### Inclusion Criteria

- 1. Adult male and female ages 18-75.
- 2. Patients meeting International Headache Society criteria for migraine with and without aura.
- 3. Patients reporting 2-8 migraine attacks per month.
- 4. Patient must be able and willing to comply with the required follow-up schedule
- 5. Patient must be able and willing to provide written informed consent
- 6. Patient was not on preventive medications for at least two months

### **Exclusion Criteria**

- 1. Has other significant pain problem (e.g. cancer pain ,fibromyalgia or other head or facial disorder) that in the opinion of the investigator may confound the study assessments
- 2. Has severe cardiac or cerebrovascular disease.
- 3. Has uncontrolled high blood pressure (systolic > 160 mmHg, diastolic > 100 mmHg after 3 repeated measurements within 24 hours).
- 4. Is currently implanted with an electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagus nerve neurostimulator ,deep brain stimulator, spinal stimulator, bone growth stimulator cochlear implant, Sphenopalatine ganglion stimulator or Occipital nerve stimulator).
- 5. Known epilepsy.



Protocol number: TCH-003 

- 6. Use of Cannabis including medical use.
- 7. Has chronic migraine (more than 15 headache days per month).
- 8. Has undergone nerve block (occipital or other) in the head or neck within the last 2 months.
- 9. Has received Botox injections within the last 6 months.
- 10. Is pregnant or thinking of becoming pregnant during the study period, or of childbearing years and is unwilling to use an accepted form of birth control.
- 11. Is participating in another clinical study in Migraine treatment or prevention.
- 12. Does not possess the basic cognitive or motor skills needed to operate android cell phone.

### **Study Procedures**

Potential patients signed informed consent prior to any study procedure. The patient medical history, migraine history, use of concomitant medications and diagnosis were recorded. Patients found eligible by meeting all the inclusion criteria and none of the exclusion criteria received documented training whereupon its successful completion the investigational device was provided to study participants for home use.

As per the instructions for use, participants were instructed to activate the device at the onset of a migraine attack and manually adjust stimulation intensity to a level where it is perceivable but not painful. Patients were requested to refrain from use of rescue medications prior to and during the first two hours following treatment by the device, and if they could not comply with this, record medications usage in the smartphone application.

Five 20-minute long stimulation protocols were programmed into each unit; four active programs at 100-120 Hz, with primary phase widths of 200 (P200), 150 (P150), 100 (P100) and 50 (P50) microseconds, and one placebo stimulation protocol (P0) at 0.1 Hz frequency with 45 microseconds long pulses. Stimuli were given at random sequences with the following distribution: P0 and P200: probability of 1/3 each, P50, P100, P150: probability of 1/9 each. Randomized sequences of programs were generated independently for each participant.

Both patients and study personnel were blinded to the order of individual treatments.

Via the smartphone application, each participant was asked to rate his/her migraine pain level four times using a Numeric Pain Rating Scale (NPS, values 0-10): (1) upon starting the treatment, (2) during (halfway through treatment program), (3) at the end of treatment, as well as (4) two hours after treatment.

At the beginning of each treatment, participants were asked to provide feedback using the application regarding the time elapsed from start of migraine attack to start of the treatment. In case of failure to provide feedback regarding pain level post-treatment, telephone follow-up was performed by study investigator staff to solicit such feedback. Follow up phone calls were performed to record changes in medical condition, concomitant medication, migraine therapy and adverse effects. Unscheduled visits were recorded, and termination visit were scheduled upon the completion of the study as defined by a maximal number of 20 complete treatment cycles but no longer than 6 months from enrollment. (whichever is fulfilled first). In the event of premature discontinuation an early discontinuation visit was scheduled. End of study interview




was performed soliciting feedback regarding device usability, burden of treatment, use of migraine medications during the study period, as well as free comments.

### **Study Endpoints**

- The primary efficacy endpoint of the study was the proportion of responders, where a responder is defined as subject with clinically significant decrease in pain score measured by Numeric Pain Rating Scale (NPS) of at least 50%, 2 hours post treatment as compared to baseline in at least 50% of treatments.
- The second primary performance endpoint was relative pain reduction at 2 hours post treatment as compared to baseline.
- The primary safety endpoint was evidence of device related adverse effects.

Burden of treatment was assessed by mean scores of post-study questionnaire. Success was defined as superior performance of active treatments as compared to sham treatment. The protocol provided for enrollment of up to 100 patients.

### **Summary of Results**

The pilot study was performed between June 2015 and March 2016. A total of 86 participants were provided with the Nerivio Migra devices for use as part of this clinical study.

A summary of participants' demographic characteristics is presented in **Table 2** below.

| | Female | Male |
|---|---|---|
| N (%) | 69 (80%) | 17 (20%) |
| Age mean (min-max, STD) | 45.2 (22-72, 11.7) | 48.8 (26- 67, 11.7) |
| Migraine attacks per month, mean (STD) | 5.1 (2.7) | 5.34 (2.3) |
| Mean pain intensity during attack | 8.9 | 8.6 |
| Occurrence of aura | 40 (58%) | 11 (65%) |

Table 2 – Pilot Study Population

Seventy-two participants successfully treated at least one migraine attack. The remainder of participants either did not treat their attacks per protocol, or failed to provide complete feedback. One participant was excluded from statistical analysis due to repeated use of rescue medications concurrently with the electro stimulation treatments. Complete reporting was obtained for 70% of activations for P200, P150, P100 programs, 58% of activations of P50 and 28% of placebo activations.

No adverse events related to the device and no side effects were reported.

Observed outcome measures based on ITT analysis are summarized in **Table 3** below.

| Sham | Active programs |
|------|-----------------|




| | PO | P200 | P150 | P100 | P50 | Overall active programs (p vs. placebo) |
|---|---|---|---|---|---|---|
| %50% (%<br>responders), N=71 | 26% | 46%<br>(0.04) | 48%<br>(0.06) | 39%<br>(0.4) | 44%<br>(0.14) | 64%<br>(significance level 0.005) |
| Relative pain reduction (%) | -2 | -20<br>NS | -26<br>P=0.02 | -16<br>NS | -18<br>NS | Model p=0.031 |
| Pain grade<br>reduction (%<br>responders), N=57 | 24% | 58%<br>(0.02) | 52%<br>(0.08) | 40%<br>(0.44) | 48%<br>(0.20) | 76%<br>(significance level 0.005) |
| No pain after two<br>hours (%<br>responders), N=57 | 6% | 30%<br>(0.004) | 12%<br>(0.56) | 23%<br>(0.06) | 26%<br>(0.14) | 44%<br>(significance level 0.005) |

### Table 3 – Pilot Study Results

Our results show that remote electrical stimulation allowed to achieve significant reduction in the migraine pain. Analysis per pain grades, as has been used for triptans, shows results similar to the triptans per pain reduction and pain elimination. When taking all active stimulation protocols together, 64% of the patients had more than 50% pain reduction, in more than half of their treated attacks. Relative pain reduction for the active stimuli ranged between 16 and 26%, while for the placebo stimulation the reduction was of 2% only. Mean pain level at device activation point was 4.6. Overall ANOVA based effect was significant (p=0.031), with significant effect in post hoc analyses for the P150 protocol.

In terms of change in pain grades, reduction from moderate or severe to mild or none was reported by 58% of the participants in response to the strongest stimulation program (P200, widest pulse), as opposed to 24% for placebo. Overall, 76% of subjects reported such reduction to active stimulation (significant at 0.005 level vs. placebo). Reduction to no pain outcome occurred in more than 50% of activations for 30% of participants when the strongest program was activated, as opposed to 6% for placebo. In the course of the study, 64% of participants who provided feedback on at least one active program activation reported at least 50% pain reduction in more than half of their activations and are considered responders to the evaluated treatment. This is significantly higher than the 26% responder to placebo activations (p=0.005).

In the end-of-trial interviews, subjects indicated (i) Reduction in amount of migraine medications during study period (mean questionnaire score was 1.5, where 1 means "same amount", 2 means "less"); (ii) overall burden of treatment was considered very low – mean score was 2.5 (between "neutral" and "not at all"); and (iii) the device and application were found easy to use by a majority of study participants (mean questionnaire score was 3.85 (between "easy" and "very easy")).




# 4.3 Clinical Investigation Risks and Benefits

### 4.3.1 Anticipated Benefits

Sponsor's pilot study demonstrated a significant effect of Nerivio Migra in alleviating migraine pain (see pilot study results above). It is anticipated that patients will experience similar effect under the setting of the current study.

Another known benefit to patients participating in such a study is the ability to learn more about their medical condition through the assessments that will be performed throughout the course of the study. Additionally, patients will be closely observed by the study staff throughout their participation in the study. Last, all assessments associated with the study, as well as the study device, are provided at no charge to the participants.

#### 4.3.2 Risks and Adverse Effects

Technical characteristics and electrical output of Nerivio Migra device are similar to other known and approved for personal use TENS devices applying electrical stimulation for pain relief purpose (see Table 1). Safety of the Nerivio Migra has been extensively tested and confirmed through bench performance testing (see section 3.5.1) as well as throughout sponsor's pilot clinical study with the device. No device related adverse events were recorded in the course of the pilot study, and treatment was well tolerated by participants.

Current study design does not require application of electrical stimulation for unusually prolonged periods, or other circumstances where the use of the device has not yet been validated. Hence this protocol presents minimal risks to the subjects and adverse events are not anticipated beyond those reported for other TENS devices. Potential expected device side effects are listed in section 14.7.

No information is available for use of the Nervio Migra and pregnancy. Thus, women who are pregnant are not eligible for inclusion in this study.

As discussed with the FDA at a Pre-submission meeting (September 2016), the Nerivio Migra is accepted as a Non-Significant Risk (NSR) device and the proposed clinical study meets the criteria of a Non-Significant Risk (NSR) device study.

### 4.3.3 Risk Control and Mitigation

The following efforts will minimize risks to patients in the study:

- Conduct of the study following successful completion of extensive bench performance testing and careful risk analysis.
- Selection of investigators who are experienced and skilled in management of patients with migraine.
- Clearly defining the inclusion and exclusion criteria such that only appropriate patients are enrolled in the study.




- Establishment of a training program for study staff members (investigators and coordinator) and use of tools that will ensure proper training to the patients for home use of the device.
- Maintaining a support team (e.g. technician, call center for massages, etc.) to assist the sites and coordinators.

#### 4.3.4 Risk-to-Benefit Rationale

The sponsor believes that the Nerivio Migra device holds great potential to provide an efficient and low risk treatment option to the population of migraine sufferers. Assessing the risks against the potential benefits of the use of the Nervio Migra for alleviating migraine pain, sponsor and the principal investigators (PIs) have determined that there is a high likelihood that the expected benefit may outweigh the risk in patients fulfilling the study eligibility criteria.




## **5 OBJECTIVES & HYPOTHESES**

# 5.1 Objective

To demonstrate the safety and effectiveness of the Nerivio Migra electro stimulation device for the reduction of migraine headache during an attack of migraine with or without aura.

# 5.2 Hypothesis

Electro stimulation delivered transcutaneously to the peripheral nervous system at onset of a migraine attack significantly alleviates headache pain demonstrated by a significant difference between proportions of responders to the active treatment stimulation and the sham control without unexpected device related adverse effects.



Protocol number: TCH-003


### 6 DESIGN OF THIS CLINICAL STUDY

### 6.1 Description

This is a prospective, randomized, double-blind, sham controlled multi-center clinical trial to test the ability of the Nerivio Migra neuromodulation device to relieve the patient's migraine pain during a migraine attack. The study will enroll up to 270 patients diagnosed with migraine with or without aura, per the inclusion and exclusion criteria. These patients will be individually and randomly assigned to either treatment group or control group. For sham control, electrical pulses of similar width and intensity, but much lower frequency compared to the active device will be administered. This sham program produces pulses that are perceivable by the user, thus maintaining the blinding, but on the other hand do not have therapeutic qualities, based on existing knowledge of parameters range of electro stimulation treatments [5-7, 18].

1<sup>st</sup> visit – screening, enrollment and training on the application in diary mode

Following successful screening, enrollment interview and signing of informed consent, participants will be provided with the Nerivio Migra application (either installed on their own smartphone, or on a smartphone provided by the study coordinator). The participants will be trained how to operate the application and report their migraine attacks in the patient diary mode, which is part of the application. The site personnel will be required to approve the training session in the CRF.

### Stage 1 - Roll in phase

The Roll-in is a period of 15 - 30 days in which at least two (2) and no more of eight (8) migraine attacks has been occurred. During this period, baseline information including mean frequency and severity of migraine attacks, occurrence of other headaches, presence of ICHD-3 diagnostic criteria for migraine with or without aura and use of preventive and rescue medications will be recorded.

### 2<sup>nd</sup> visit

Following the Roll-in phase, the participants will arrive to the clinic and their compliance to the study procedures and eligibility to continue to the next phase will assessed.

For the study purpose, an eligible subject for stage 2 is a subject that comply with the following criteria:

- Subject had at least 2 and no more than 8 migraine attacks during the Roll in stage
- Migraine attacks were reported as required by the protocol (within 60 min from onset, complete reports at t=0 and t=2 hours) in at least the following attacks percentage:
  - o 1 out of 1 attack (100% compliance)
  - o 2 out of 2 attacks (100% compliance)
  - o 2 out of 3 attacks (67%% compliance)
  - 3 out of 4 attacks (75% compliance)
  - 4 out of 5 attacks (80% compliance)
  - o 5 out of 6 attacks (83% compliance)
  - o 6 out of 7 or 8 attacks (75-85% compliance)




Participants that will be eligible to continue to the treatment phase will undergo the following:

- Participant will be randomized into one of the two study group (Active or Sham device)
  Investigational devices will be programmed in active or sham mode with a 1:1 ratio, in
  order to achieve the desired ratio between active and control groups sizes, stratified with
  by use of preventive medications.
- 2. Participant will be trained on the device, the application (in diary and treatment modes), the treatment procedures and the key elements critical for the success of the study:
  - Apply the Nerivio Migra as soon as possible following the onset of the migraine symptoms and NO LATER than 60 min from onset
  - Refrain from taking any rescue medication 2 hours following the start of treatment.
  - Perform the treatment for a period of at least 30 minutes (recommended treatment time is 45 minutes).

During the training for the treatment phase, participants will operate the device and the appropriate intensity range for each individual participant will be defined with the study team in a way that the treatment stimulation is "well-perceived but not painful" for the participant. This individual Intensity level will be recorded, and the participant will be asked to operate the device within this range as a default.

If the research staff recognizes during the training that the patient cannot tolerate the feeling of the electrical stimulation, the patient will be withdrawal from the study, as described in section 6.5.7 patient withdrawal criteria.

### Stage 2 - Parallel arms, double- blind treatment phase.

Participants will be instructed to activate the device at onset of a qualifying migraine attack and manually adjust stimulation intensity to a level within the pre-defined range, where it is well perceived but not painful. A qualifying migraine attack shall be preceded by at least 48 hours of freedom from migraine. Patients will be requested to refrain from use of rescue medications prior to and during the first two hours after treatment with the device, and if they cannot comply with this, record their use of rescue medications (migraine specific drugs or other medications or therapies that may be used to treat pain, from a pre-specified list) in the mobile application.

Via the smartphone application, each participant will be asked to rate his/her migraine pain level three times using Pain Grades Scale (0 - no pain, 1- mild pain, 2- moderate pain, 3 – severe pain): (1) upon starting the treatment, (2) two hours after start of treatment, (3) 48 hours after start of attack. At the start of each treatment, participants will be also asked to provide time elapsed from start of migraine symptoms to start of the treatment. Participants will be also asked to provide feedback regarding their use of medication (migraine specific drugs or other medications or therapies that may be used to treat pain, from a pre-specified list), presence of nausea, photophobi, phonophobia or allodynia, and treatment perception. After providing feedback at two hours after start of treatment and in case of pain recurrence, participants will be allowed to re-treat the attack using Nerivio Migra device.

Adverse events will be reported.



For the purpose of the study endpoints analysis, the following treatments will be considered for both active and placebo groups:

- The 1<sup>st</sup> reported treatment in the double-blind treatment stage will be considered as a "run-in test" treatment, to assess the patient competence to activate the device and report his migraine headache level at the required time periods. This treatment will be included in the safety endpoint analysis only. It <u>WILL NOT</u> be included in any of the primary and secondary performance endpoints analysis.
- The 2<sup>nd</sup> reported treatment (1<sup>st</sup> after the "run-in test" treatment) will be considered as a valid treatment and will be used for the analysis of the primary performance endpoint, as well as for the secondary, exploratory and safety endpoints, as defined in section 6.3.
- The subsequent treatments (3<sup>rd</sup>, 4<sup>th</sup> and 5<sup>th</sup> treatments if performed) will be considered as valid treatments and will be used for the "repeatability" exploratory endpoint analysis and the safety endpoint analysis, as defined in section 6.3.

Duration for each patient will be approximately two months – up to one month of roll-in stage followed by treatment stage of up to five qualifying attacks (with the first reported attack considered as a" run-in test" (pilot) treatment, while the following four reported attacks considered as valid treatments for endpoint analysis) over the course of one month (whichever is achieved first). An optional open-label extension of two months is available.

Post study questionnaire will include patient global impression of change [27], blinding and usability assessments.

Study flow is schematically presented in **figure 6** below.






Figure 6. - Study Design

#### 6.2 Measures to Minimize Bias

A number of measures are built into the study design and procedures in order to minimize various potential sources of bias.

Implementation of the 2-4 weeks of roll-in period in conjunction with baseline assessment (questionnaire) mitigates <u>recall bias</u> and allows more reliable assessment of baseline headaches frequency, duration and severity.

<u>Gender selection bias</u> will be eliminated due to recruiting patients in headache clinics, emergency and neurology departments.

Randomization is employed to avoid bias in participants' allocation to study arms.

Double blind design is ensuring collection of bias free efficacy data. Specific measures will be taken to ensure blindness (refer to Section 6.2.2).

Participants will define their intensity working range during the training session, prior to treatment phase, to ensure that the intensity level is the appropriate level they require and tolerate.

Detailed statistical analysis plan will be developed prior to study start to mitigate <u>interpretation</u> <u>bias</u>.




#### 6.2.1 Randomization

Randomized allocation of active and sham devices with stratification to use of preventive medications will be performed. Every site will be allocated a stock of identically looking, numbered devices of both kinds.

## 6.2.2 Procedures to ensure blinding

This is a double-blind study: neither the patient, nor the investigators will be aware of arm allocation of each study participant. Maintaining double blind design is a known challenge in non-invasive neuromodulation devices trials. Several means are planned to ensure the double-blind aspect of this trial.

- Selection of identically looking, active sham devices as control means is only a single step aimed at maintaining blindness.
- Adherence to randomization procedure by clinical staff is critically important.
- Importance of adherence to study design and procedures will be explained to participants in the course of enrollment.
- No information regarding expected stimulation perception will be provided, except for the fact that stimulation intensity adjustment control will allow to adjust intensity to a "well perceived but non-painful" level.
- In order to achieve blinding, participants will be trained individually. A training clip will be used for training, in order to minimize staff exposure to participants' reaction to and tolerability of treatment intensity.
- In the course of the trial, participants will not be asked directly any questions regarding treatment perception.
- The clinical staff will be instructed to not engage in any discussions regarding anticipated treatment perception.

End of study questionnaire will include individual blinding assessment to examine whether the blinding was well maintained throughout the study.

# 6.3 Study Endpoints

#### 6.3.1 Primary Endpoint

#### Reduction of Migraine Headache:

The proportion (%) of patients reporting reduction in their pain level 2 hours post-treatment without rescue medications from severe or moderate to mild or no pain, or from mild to no pain in their first treated migraine attack (excluding the "run-in test" treatment).

For calculating this endpoint, only the 1<sup>st</sup> reported treatment following the "run-in test" treatment will be used.



Protocol number: TCH-003


#### 6.3.2 Secondary Endpoints

#### Secondary Performance Endpoints

#### 1. MBS Relief:

Proportion (%) of patients reporting, 2 hours post-treatment, freedom from their most bothersome migraine-associated symptom (MBS) other than a headache, in their first treated migraine attack (excluding the "run-in test" treatment). MBS may be nausea, photophobia, phonophobia or allodynia – as defined by each subject.

#### 2. Migraine Headache Relief AND MBS Relief:

Proportion (%) of patients reporting 2 hours post treatment response to both the primary and the first secondary endpoints.

#### 3. Pain-free at 2 hours:

The proportion (%) of subjects reporting freedom from migraine pain at 2 hours post-treatment without medications in their first treated migraine attack (excluding the "run-in test" treatment)

#### **6.3.3** Exploratory Endpoints:

1. Sustained pain-free 48 hours with single use of the device:

The proportion (%) of subjects reporting pain-free at 2 hours, and no return of any pain or use of rescue/acute medication, or reuse of device between 2 hours and 48 hours, in their first treated migraine attack (excluding the "run-in test" treatment).

2. Sustained Headache Reduction for 48 hours with single use of the device:

The proportion (%) of subjects reporting treatment response 2 hours post-treatment without rescue medications, and no return to baseline level of pain at time of treatment, or use of rescue/acute medication, or reuse of device between 2 hours and 48 hours, in their first treated migraine attack (excluding the "run-in test" treatment).

Treatment response is defined as:

- pain level reduction from moderate or severe at baseline to mild or none, OR:
- pain level reduction from mild to no pain.
- 3. Sustained pain-free 48 hours with reuse of device

The proportion (%) of subjects reporting pain-free at 2 hours, and no return of any pain or use of rescue/acute medication except for reuse of device between 2 hours and 48 hours, in their first treated migraine attack (excluding the "run-in test" treatment).

4. Sustained Headache Relief 48 hours with reuse of the device:



Protocol number: TCH-003


The proportion (%) of subjects reporting Treatment Response at 2 hours, and no return to baseline level of pain at time of treatment, or use of rescue/acute medication except for reuse of device between 2 hours and 48 hours, in their first treated migraine attack (excluding the "run-in test" treatment).

Treatment response is defined as:

- pain level reduction from moderate or severe at baseline to mild or none, OR:
- pain level reduction from mild to no pain.
- 5. Sustained relief of MBS with a single use of the device

The proportion (%) of subjects reporting freedom from MBS at 2 hours, and no return of MBS, or use of rescue/acute medication between 2 hours and 48 hours, in their first treated migraine attack (excluding the "run-in test" treatment).

6. Sustained relief of the MBS with reuse of the device:

Proportion (%) of patients reporting, 48 hours post the first treatment, freedom from their most bothersome migraine-associated symptom other than headache (MBS), possibly with reuse of the device, in their first treated migraine attack (excluding the "run-in test" treatment).

7. Within-patient consistency of the primary endpoint in subsequent treatments:

The repeatability of migraine headache reduction, as described in the primary endpoint definition, in subsequent treated attacks.

Thus, this endpoint measures the % of patient responding to the primary endpoint in at least 50% of their treated attacks (excluding the "run-in test" attack)

#### 6.3.4 Safety Endpoints:

- Adverse events related or unrelated to the study device.
- Treatment tolerability

# 6.4 Methods and Timing of Assessing, Recording and Analyzing Variables

Data capture and management are described in detail in the Data Management Plan. List and structure of individual eCRFs are also given in the Data Management Plan. Data monitoring procedures are described in detail in the study's Monitoring plan. The study will rely to a large degree on electronic data capture methods.

## 6.4.1 Types of Data

Overall, data collected in the course of the study may be divided into three categories:




- captured by clinical personnel. This includes demographic characteristics, baseline
  migraine parameters, end of study questionnaires, adverse events reports. Source data
  may be paper worksheets, further transferred into eCRFs maintained by the EDC system.
- 2. patient reported outcomes. This includes feedback entered via the smartphone application regarding migraine pain level, migraine symptoms, treatment perception, rescue medications. These data are used for calculation of study endpoints. Here, source data will be electronic, followed by automatic transfer to eCRFs.
- 3. additional information and technical data, captured by means of a system of log files by the Application. This includes stimulation activation times, applied stimulation intensity, device defects information, and other.

## 6.4.2 Clinical Study Variables and Data Capture Tools

This section provides an overview of collected PRO data and its capture tools.

#### 6.4.2.1 Start attack/episode PRO feedback data

The screen provides for collection of the following data:

| | D | Control | Wil and the second |
|---|---|---|---|
| Item | Description | Control type | Values range |
| Current migraine | Current | Dropdown list | Mild (1), |
| pain level | migraine pain | | Moderate (2), |
| | level in pain | | Severe (3). |
| | grade categories | | |
| Time from onset | Time from onset | Dropdown list | 1) Within 30 minutes |
| of migraine pain | of migraine pain | | 2) Between 30 to 60 minutes |
| | | | 3) 60 minutes or more |
| Nausea | Presence of | Radio buttons | Y/N |
| | nausea | | |
| Sensitivity to | Presence of | Radio buttons | Y/N |
| light | photophobia | | |
| Sensitivity to | Presence of | Radio buttons | Y/N |
| sound | phonophobia | | |
| Increased skin | Presence of | Radio buttons | Y/N |
| sensation | allodynia | | |
| MBS | Most bothering | Dropdown list | 1) Nausea |
| | symptom (other | | 2) Photophobia |
| | than headache) | | 3) Phonophobia |
| | | | 4) Allodynia |




#### 6.4.2.2 2h PRO

This feedback dialog appears 2h after the treatment program has started.

The screen provides for collection of the following data:

| Item | Description | Control type | Values range |
|---|---|---|---|
| Current<br>migraine pain<br>level | Current migraine pain level in pain grade categories | Dropdown list | No pain (0), Mild (1), Moderate (2), Severe (3). |
| Medication | Whether rescue<br>medication was<br>taken within 4h<br>prior treatment<br>until the 2h<br>follow-up period. | Radio buttons | Y/N |
| Medication time | If patient indicates taking medication, she needs to insert the time when medication was taken | Dropdown list | <ol> <li>Before start of treatment</li> <li>Less than 2 hours after start of treatment</li> <li>2 hours or more from starting the treatment</li> </ol> |
| Medication name | Rescue<br>medication | Dropdown list | From a pre-defined list |
| Nausea | Presence of nausea | Radio buttons | Y/N |
| Sensitivity to light | Presence of photophobia | Radio buttons | Y/N |
| Sensitivity to sound | Presence of phonophobia | Radio buttons | Y/N |
| Increased skin sensation | Presence of allodynia | Radio buttons | Y/N |

#### 6.4.2.3 48h PRO

The screen shall provide for collection of the following data:

| Item | Description | Control type | Values range |
|------|-------------|--------------|--------------|



Protocol number: TCH-003 

| Current<br>migraine pain<br>level | Current<br>migraine pain<br>level in pain<br>grade categories | Dropdown list | No pain (0), Mild (1), Moderate (2), Severe (3). |
|---|---|---|---|
| Medication | Whether rescue<br>medication was<br>taken within the<br>last 46h | Radio buttons | Y/N |
| Medication name | Rescue<br>medication | Dropdown list | From a pre-defined list |

# 6.4.3 Methods and Timing of Assessing, Recording and Analyzing Variables

Once the last patient will have completed the study and all the queries have been resolved, database will be locked, cleaned and exported for final statistical analysis. Study report will be issued following final database lock.

Only data from the first 2h of the 1<sup>st</sup> treated migraine attack following the "run-in test" attack will be used for analysis of the study **primary** endpoint. A new migraine attack is an attack that that had a "freedom from pain" period of at least 48 hours prior the attack.

Recurrent treatments within 46 hours from first treatment of an attack are allowed, and are collected as exploratory data. Use of rescue medication within the 48 hours from start of 1<sup>st</sup> treatment of the attack is considered a failure for sustained relief assessment.

#### 6.4.4 Data Flow and Management

Data management function will be supported by a cloud based EDC system developed by Clear Clinica (Modi'in, Israel). Clear Clinica provides services for collection and remote monitoring of clinical trials data, compliant with HIPAA and 21 CFR Part 11.

EDC portals with secure authorized access will be made available to every participating site, as well as to the study monitor.

Data captured by clinical personnel will be entered directly into pre-specified eCRF screens by site personnel. Data from paper sources will be entered into the study database. Automatic data checks will be implemented for majority of entry fields to provide opportunity for resolving data inconsistencies as close as possible to real time. Effort will be made to identify missing or incorrect data and resolve the issues promptly.

Data collected onto the smartphone application will be directed to a secure cloud based database where it will undergo analysis aimed at detection of missing data and other inconsistencies. The smart phone will transmit PRO and technical data containing activation times, stimulation intensity and ePRO via the smartphone to a central electronic database for analysis. Activities



Protocol number: TCH-003 

such as repeatedly aborted programs, missing feedbacks, inconsistent stimulation intensity adjustments, and similar, will be communicated to research coordinator of the corresponding site, using participants' ID codes. Automated means were developed to identify and provide corresponding notifications regarding events that may lead to protocol deviations and/or missing data, and which resolution may require involvement of study staff. Examples of such events include missing PRO data or low device battery level. An automated system was implemented to notify the participant, site study coordinator and Sponsor study monitor on the above events. Missing data will be identified automatically by a script running on Clear Clinica's cloud, and queries will be generated to participants and corresponding site study coordinator. Near real time detection of problems in accumulating data will allow timely generation and resolution of queries. Intermediate data processing and translation into eCRF format are performed at this stage. Processed data are further pushed into the EDC system.

Schematics of data flow are presented in **figure 7**.



Figure 7. - Schematics of data flow




Back-up of the database is performed daily. In addition, copy of each participant's ePROs and other activity is stored in his/her smartphone memory and can be retrieved in case such need occurs.

Study database will be locked and exported using EDC tools into SAS compatible format for interim and final statistical analyses.

Query resolution will be performed using EDC tools.

All paper based source data and relevant medical documents meant to serve also as source documents will be maintained by the sites and available as eCRF attachments. Patient identification will be blackened from all data. Patients will be identified by their codes. The site investigator is responsible for ensuring that eCRFs are filled in a timely manner and relevant paper documents are properly stored. Investigator will provide the documents to the sponsor either through the sponsor representative or by mail per sponsor request.

Access to data will be authorized and controlled, in accordance with relevant laws and guidelines.

Study will be performed according to the protocol. At each site, the PI will appoint staff member(s) that will be responsible for completing the Case Report Forms supplied by the sponsor.

Specifics of data query handling are given in Data Management and Monitoring plans.

Audit trail for data entry and corrections will be maintained.

# 6.4.5 Procedures for Review of Data

A detailed description of data queries, their resolution and overall data flow can be found in the Data Management Plan.

Missing PRO data will be identified by a dedicated software running on the cloud closely to real time. Corresponding queries will be issued to study participants and site study coordinator. Effort will be made to resolve such queries as close as possible to real time.

# 6.4.6 Data Monitoring Committee

An independent Data Monitoring Committee (DMC) is charged with the task of providing regular oversight of the data monitoring issues as detailed in the document: "DMC". These experts will periodically review and evaluate the accumulated data for study progress. The DMC will make recommendations concerning continuation, modification, or termination of the study. The Data reviewed by the DMC will include a summary of the following topics:

- <u>Study progress</u>: Subject recruitment, comparison with targeted recruitment, retention, protocol adherence, and quality of data collection procedures.
- Treatment Monitoring: Data on treatment integrity and adherence.
- <u>Safety Monitoring</u>: Data related to the safety of the subjects, including any adverse events or side effects related to the treatment.
- <u>Efficacy monitoring</u>: Interim efficacy analysis is to be performed per algorithm presented in Section 7.6.



Protocol number: TCH-003 

• Futility monitoring: Futility will be assessed at the time of interim analysis.

## 6.4.7 Total Expected Duration of the Clinical Investigation

The anticipated duration of the study is up to 12 months.

## 6.5 Subjects

#### 6.5.1 Inclusion Criteria

Patients need to fulfill all the below Inclusion criteria:

- 1. Subject is 18-75 years old.
- 2. Subject meeting the ICHD-3 diagnostic criteria for migraine with or without aura
- 3. Subject reporting 2-8 migraine attacks per month.
- 4. Stable migraine preventive medications in the last two months prior to recruitment (No change in usage or dosage).
- 5. Subject must be able and willing to comply with the protocol
- 6. Subject must be able and willing to provide written informed consent

#### 6.5.2 Exclusion Criteria

Patients are excluded if they have any of the following:

- 1. Subject has other significant pain, medical or psychologic problems that in the opinion of the investigator may confound the study assessments
- 2. Subject is currently implanted with an electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagus nerve neurostimulator ,deep brain stimulator, spinal stimulator, bone growth stimulator cochlear implant, Sphenopalatine ganglion stimulator or Occipital nerve stimulator).
- 3. Subject has known uncontrolled epilepsy.
- 4. Any use of Cannabis including medical use.
- 5. Subject has > 10 headache days per month.
- 6. Subject has undergone nerve block (occipital or other) in the head or neck within the last 2 weeks.
- 7. Subject is participating in any other clinical study.
- 8. The subject does not have the basic cognitive and motor skills needed to operate a smartphone
- 9. Pregnant, or trying to get pregnant
- 10. Subject is experiencing a menstrually related migraine
- 11. Received OnabotulinumtoxinA or any botulinum toxin injections for migraine within the previous month
- 12. Received parenteral infusions for migraine within the previous 2 weeks.



Protocol number: TCH-003


#### 13. Subject participate in a previous study with the Nerivio Migra 1 device

<u>Note</u> - Females of child bearing potential must have a negative pregnancy test and must be willing to use adequate contraceptive means during the study

#### 6.5.3 Contraindications

Contraindications for the use of the Nerivio Migra device include those known for transcutaneous electrical stimulation procedures. In addition to restrictions described in exclusion criteria, Nerivio Migra shall not be placed over open wounds or burns, or on irritated skin.

The Nerivio Migra is **NOT** intended for use in any other location except the upper arm.

## 6.5.4 Number of Subjects

The total number of patients to be treated in this study is up to 270 eligible patients (see section 7.6).

## 6.5.5 Expected Study Duration for Each Subject

Study duration per patient is up to 2 months for the roll-in and double-blind stages, and then, possibly another 2 months for the open label extension, if required.

## 6.5.6 Point of Enrollment

Patients are formally enrolled in the study once they are found eligible by inclusion and exclusion criteria, have signed an informed consent and received training on the use of the device. If the patient was not treated with the investigational device, the patient will be excluded from the mITT data analysis set.

#### 6.5.7 Patient Withdrawal Criteria

Patients may be withdrawn from the study by the PI or sponsor, if any one or more of the following events occur:

- The patient wishes to withdraw from the study without providing any explanation.
- Patient is lost to follow-up.
- Refusal of the patient to continue treatment and/or follow-up observations.
- Serious adverse event.
- Subjects who have problems/difficulties with the Investigational Product (IP) and cannot handle it independently (e.g. cannot tolerate the treatment, cannot operate the application).
- Significant protocol deviation/violation or noncompliance, either on the part of the patient or investigator.
- Decision made by the investigator that termination is in the patient's best medical interest.




- Device failure.
- Other ethical or clinical considerations upon investigator discretion.

## 6.5.8 Handling of Withdrawals

In accordance with the Declaration of Helsinki, a patient has the right to withdraw from the study at any time, for any reason, without prejudice to any future medical care by the physician or the institution. The investigator and the sponsor also have the right to withdraw patients from the study in the event of serious adverse events, protocol departures (deviations, violations and exemptions), or other reasons. Should a patient (or the patient's legally authorized representative) decide to withdraw, all efforts will be made to collect and report the next visit observations, and the reasons for withdrawal, as thoroughly and timely as possible.

Withdrawals will be recorded, analyzed and reported to local ethical committee according to local regulations.

## 6.5.9 Patient lost to follow-up

If a patient does not show for end-of-study visit and cannot be contacted to collect follow-up information, he/she will be counted as a 'missed visit'. Prior to counting the patient as a 'missed visit' the following will be performed:

- Repeated, documented attempts to contact the patient via all available means.
- Repeated, documented attempts to contact the patient's general practitioner or referring physician.
- If a visit cannot be arranged, obtain as much information as possible through all communication means with the patient and/or his/her treating physician.

If a patient is lost to follow-up, the methods used to attempt to contact the patient should be noted. At least three attempts should be made to contact the patient and/or his/her treating physician via all available routes, and a certified letter should be sent to the permanent address on file.

#### 6.5.10 Enrollment Period

The anticipated enrollment rate is expected to be approximately 6-10 patients per month, depending on participating site. Enrollment period is expected to be up to six months long.

# 6.5.11 Procedures for Replacement of Subjects

No subject replacement is planned.




## 6.6 Study related Procedures

#### 6.6.1 General

The potential candidates will be screened to assess whether they are appropriate candidates for inclusion in this study. Informed consent will be obtained prior to initiation of any of the following clinical procedures that are performed solely for the purpose of determining eligibility for research. Pregnancy test for female patients with childbearing potential will be performed. The patient medical history, migraine history and diagnosis will be recorded and verified, the use of concomitant medication will be recorded in designated case report forms. Eligible patients will receive a documented training, and upon its successful completion the application will be installed on the participant's phone (or on a dedicated phone supplied by the Sponsor, depend on participant's request) during the 1st phase. Investigational device will be handed to study participants for home use prior the 2<sup>nd</sup> phase. As per the IFU, participants are instructed to activate the device at the onset of a migraine attack and manually adjust stimulation intensity to a level where it is perceivable but not painful, as defined during the Randomization/training visit. Participants are requested to refrain from use of rescue medications prior to and during the first two hours after treatment and, if could not comply with this, record their use in the cellular application. Via the smartphone application, each participant will be asked to rate his/her migraine pain level three times: (1) upon starting the treatment, (2) two hours after treatment, (3) 48 hours after first treatment corresponding to the current migraine attack, using Pain Grades Scale (0 - no pain, 1- mild pain, 2- moderate pain, 3 – severe pain). At the end of each treatment, participants will be asked to provide feedback using the application regarding the time elapsed from start of migraine attack to start of the treatment, their use of medication. In case of failure to provide feedback regarding pain level post-treatment, telephone follow-up will be performed by study investigator staff to solicit such feedback. Additional migraine symptoms will be selfreported using the application. Follow up phone calls will be scheduled to record change in medical condition, concomitant medication and migraine therapy. Unscheduled visits will be recorded and termination visit will be scheduled upon the completion of the study as defined by treatment of four qualifying attacks over the course of one month (whichever is achieved first). In the event of premature discontinuation an early discontinuation visit will be scheduled.

#### 6.6.2 Visit and assessment schedule

The study requires up to four visits: (1) for screening and migraine diary training and (2) randomization and device treatment training (3) end of study, when the device is returned, and end of study assessment is performed If the patient chooses to continue to the open-label extension, additional visit (4) will be required.

## 6.6.3 Activities performed by sponsor representatives

It is the sponsor's responsibility to train the site staff and supply the devices in a timely manner.



Protocol number: TCH-003


It is also the sponsor's responsibility to communicate to other sites' representatives in regard to serious adverse events, device malfunctioning findings and other relevant information that may affect study operation.

## 6.7 Monitoring Plan

A detailed Monitoring Plan was developed for this study by the sponsor.

Monitoring functions will be performed in compliance with Good Clinical Practices guidelines per forth in ISO 14155 (2011). The major function of the clinical monitor is to observe and assess the quality of the clinical study and the data generated from it, and to ensure that patients' welfare is being kept.

Based on implementation of an EDC platform, remote monitoring will be possible and will be performed on a regular basis between monitoring visits. The Study Monitor/CRA will access the EDC to perform remote review of the data. Attention will be paid (but not limited to) to the following:

- Number of patients enrolled, per site.
- Timely data entry.
- Timely resolution of queries.
- AE/SAE and device deficiencies reporting in accordance with the protocol and according to the timelines, including adequate follow-up.
- Non-compliances documentation.
- Timely follow-up.
- Devices accountability

Due to utilization of integrated ePRO tools and EDC platform for data collection and management, electronic source data will be considered verified by nature of process validation and verification performed jointly by the sponsor and the EDC vendor and documented separately.

A well planned and prepared Initiation Visit will take place to address and train the site on aspects of protocol adherence and data monitoring processes.

The following monitoring visits are planned in the course of the study:

- After the Site Initiation, a monitoring visit close to the first few (3-5) subjects' enrollment.
- After the study completion by first few patients
- After completion of study by all planned patients

In cases where the monitor notices that the PI is performing not according to the protocol or relevant regulation, the monitor should notify the sponsor by means of the monitoring report, email notification or a separate report if needed (i.e. Deviation Report Form). A follow-up letter to the PI should include the key findings. Site revisiting regarding GCP and protocol adherence should be done by the monitor in case of repetitive deviations.




#### 7 STATISTICAL CONSIDERATIONS

## 7.1 Study Design and Aim

The study is designed as a prospective, randomized, double-blind, sham controlled multi-center clinical trial. The study aim is to demonstrate safety and effectiveness of Nerivio Migra electro stimulation device for the acute treatment of migraine attacks with and without aura.

## 7.2 Study Variables

## 7.2.1 Primary performance variable

The primary performance endpoint will be measured in the form of a binary variable which will be assigned the value of "1" if the subject reports such headache pain reduction without rescue medications, and "0" otherwise.

## 7.2.2 Secondary performance variables

The secondary performance endpoints will be measured in the form of a binary variable which will be assigned the value of "1" if the subject responds to each specific secondary endpoint, and "0" otherwise.

# 7.2.3 Exploratory performance variables

The exploratory performance endpoints will be measured in the form of a binary variable which will be assigned the value of "1" if the subject responds to each specific exploratory endpoint, and "0" otherwise.

In addition, patient global impression of change is measured via a questionnaire.

# 7.2.4 Safety variables

Incidence of all adverse events and complications by severity and relationship to study device.

Treatment tolerability as measured by a questionnaire.

# 7.3 Study Hypothesis

 $H_0$ : The proportion (%) of subjects reporting reduction of migraine headache at 2 hours post treatment without rescue medications from severe/moderate to mild/no-pain or from mild to nopain during the  $1^{st}$  migraine attack following the "run-in test" attack in the treated group = The proportion (%) of subjects reporting reduction of migraine headache at 2 hours post treatment without rescue medications from severe/moderate to mild/no-pain or from mild to no- in the  $1^{st}$  migraine attack following the "run-in test" attack in in the sham group.

 $H_A$ : The proportion (%) of subjects reporting reduction of migraine headache at 2 hours post treatment without rescue medications from severe/moderate to mild/no-pain or from mild to nopain in the 1<sup>st</sup> migraine attack following the "run-in test" attack in in the treated group  $\neq$  The




proportion (%) of subjects reporting reduction of migraine headache at 2 hours post treatment without rescue medications from severe/moderate to mild/no-pain or from mild to no-pain in the 1<sup>st</sup> migraine attack following the "run-in test" attack in in the sham group.

If the null hypothesis is rejected in favor of the alternative hypothesis and the proportion (%) of subjects responding to this endpoint in the treated group is greater than that of the sham group, the study will be deemed successful.

## 7.4 Sample Size Estimation

T The sample size for this study was calculated to test the null hypothesis with a chi-squared test, even though the final analysis may employ a regression model or a Fisher's exact test.

Sample sizes are calculated for both the primary and secondary endpoints to test the hypothesis with 80% power at a 5% level of significance. Sham success rate is assumed to be 32% and the sample size calculated for differences ranging between 15% and 20%.

#### Primary endpoint:

We assume that 50% of the subjects in the treatment arm will have successful reduction of migraine headache versus 32% in the sham arm. Hence, 234 evaluable subjects are required to detect this difference, 117 per group. Allowing for a ~15% drop-out rate, a total of 270 (135 treated vs. 135 sham) subjects should be enrolled in the study.

# 7.5 Definition of eligible treatment

An eligible patient for statistical analysis is a patient that complete the Roll-in phase and the treatment phase. An eligible migraine episode for analysis of primary and secondary endpoints includes the following

- The patient had at least 48 consecutive hours without migraine headache prior to treatment.
- Treatment is started no later than 60 minutes post the onset of migraine symptoms.
- Treatment lasted at least 30 (continuous) minutes.
- No pain medications were used from 24 hours prior the onset of the migraine, until 2 hours after the start of the treatment.
- The patient completed and reported the post 2-hour treatment questionnaire through the application.

## 7.6 Interim Analysis

An interim analysis will be performed when approximately 20-30% of the subjects reach the primary endpoint. An independent committee will review the results and recommend whether the study should be stopped for futility or continue. Details of the interim analysis will be specified in a statistical analysis plan prior to study initiation.



Protocol number: TCH-003

Page **54** of **94** 

#### 7.7 Randomization

Subject will be randomly allocated (with a 1:1 ratio) to one of the following 2 treatment groups based on a randomization scheme using the permuted block method stratified by preventive medications use and center:

- Sham Control
- Nerivio Migra group

The randomization scheme will be prepared by the study statistician using the SAS (version 9.4.) random number procedure. The block size will be fixed, and study personnel will be blinded to the randomization block size.

## 7.8 Analysis sets

#### Analysis Sets:

1. Intent to Treat analysis set (ITT)

The ITT analysis set includes all patients who are randomized and treat at least one attack.

2. Modified Intend to Treat analysis set (mITT)

The mITT analysis set includes all patients who are randomized and treat at least one attack (excluding the "run-in test" attack) within 1 hour from the attack onset.

3. Per-Protocol analysis set (PP)

The PP analysis set includes patients who are randomized and treat at least one attack (excluding the "run-in test" attack), which conforms with the protocol instructions:

- Treatment starts within one hour from attack onset.
- No rescue medication (or pain medication) is consumed within the 2 hours after start of treatment.
- The treatment is not aborted prematurely (i.e., before the first 30 minutes).
- No Pain medication 24h prior migraine onset

#### Statistical Analysis of Analysis Sets:

The ITT analysis set will serve as the main set for safety assessments

The mITT analysis set for all performance assessments.

The primary and secondary performance assessments will also be performed on the PP analysis set as a sensitivity analysis.



Protocol number: TCH-003


# 7.9 Statistical Analyses – (TBD)

Amendments to the statistical analyses section will not require IRB approval, unless driven by protocol or study design change. In that case a standalone SAP will be prepared prior to data lock for each analysis milestone.

#### 7.9.1 General Considerations

Statistical analyses will be performed using SAS® v9.4 (SAS Institute, Cary NC, USA).

All statistical tests will be two-sided. The required significance level of findings will be equal to or lower than 5%, nominal p-values will be presented. Where confidence limits are appropriate, the confidence level will be 95%.

Continuous variables will be summarized by a mean, standard deviation, minimum, median and maximum, and categorical variables by a count and percentage. For comparison of means (continuous variables), the two-sample t-test or the Wilcoxon rank sum test will be used as appropriate. For comparison of proportions (categorical variables), the Chisquared test or Fisher's exact test will be used as appropriate.

If multiple measurements are taken in a single patient, statistics described below will be appropriately modified to accommodate the within patient correlation.

# 7.9.2 Significance levels and handling of type I error

### 7.9.2.1 Type I Error

The overall significance level for this study is 5% using two-tailed tests, except for treatment by site interaction that will be tested at a significance level of 10%.

# 7.9.2.2 Hierarchy Approach for Secondary Endpoints Analysis

The hierarchy approach will be adopted for the primary and secondary endpoints to control type I error due to multiple endpoint testing. Thus, the primary endpoint will first be analyzed and only if p<0.05, will the secondary endpoints be analyzed.

# 7.9.3 Demographic and Other Baseline Characteristics

Demographic and baseline condition related characteristics will be tabulated and compared between the study groups by data type. Continuous variables will be summarized by a mean, standard deviation, minimum, median and maximum, and categorical variables by a count and percentage.

This data will include:

- Demographic data
- Medical history
- Migraine preventive medication
- Other concomitant medication




- Migraine attacks characteristics per ICHD-3 diagnostic criteria for migraine with and without aura
- Physical examination
- Laboratory (pregnancy) tests for women of childbearing potential

## 7.9.4 Disposition of Patients

The numbers of patients who entered the study and completed each stage of the study will be provided per month, as well as the reasons for all post randomization discontinuations, grouped by major reason, e.g., lost to follow-up, adverse event, poor compliance, did not administer any treatment (with reasons). A list of discontinued patients, protocol deviations, and patients excluded from the performance analysis will be provided as well.

## 7.9.5 Performance Analyses

#### **Primary performance:**

A count and percentage of subject treatments responding to the primary performance endpoint will be calculated and presented for both study groups each with a two-sided 95% exact confidence interval. The groups will be compared with a chi-squared test, and a Fisher's exact test.

If the null hypothesis is rejected in favor of the alternative hypothesis and the proportion (%) responders in the treated group is greater than that of the sham group, the study will be deemed successful.

The primary endpoint will also be evaluated stratified by center using a Mantel-Haenszel test to assess the center by group interaction.

A sensitivity analysis of the primary endpoint will be performed to assess the impact of missing data on the study outcome. This will be performed using several possible imputation methods. A subject who took rescue medication during the 2 hours post treatment is considered as being in pain. The PP analysis will be performed without these attacks.

Adjustment for other covariates such as demographics or other baseline patient characteristics may be performed by adding these variables into a logistic regression model.

Subgroup analysis according to use of preventive medications, time from onset of attack till treatment and intensity of stimulation will be performed and reported by adding these variables to a logistic regression model.

#### <u>Secondary performance</u>:

The secondary performance variables will be summarized by a count and percentage and compared with a chi-squared test.

#### **Exploratory performance:**



Protocol number: TCH-003


A count and percentage of patients responding to each of the exploratory performance endpoints will be presented. The groups will be compared with a chi-squared test and a Fisher's exact test.

Patient global impression of change (total score) will be summarized by descriptive statistics per treatment group and compared between the groups with a t-test.

Frequency of use of rescue medication will be summarized by descriptive statistics per treatment group and period (roll-in vs. treatment) and compared between the groups with Poisson regression.

## 7.9.6 Safety Analysis:

The primary safety variable, the cumulative incidence (and 95% CI) of device related adverse events (AEs) throughout the study, will be presented in tabular format and will include incidence tables by severity.

Adverse event rates will be compared between the study groups with a Fisher's exact test.

Serious adverse events will be listed and discussed individually.

Treatment tolerability will be compared between the study groups, the number and percent of subjects who fail to complete the study and the number and percent of subjects who fail to complete the study because of Adverse Events will be presented as well

# 7.9.7 Handling of Missing Data

A sensitivity analysis of the primary end-point will be performed to assess the impact of missing data on the study outcome using possible imputation methods for binary data. A "worse case" scenario analysis will be performed as well where subjects with missing data for the binary response assessment will be considered as a non-responder/ non-success.

Imputation of missing data may be performed on secondary and exploratory endpoints as well.

# 7.10 Pooling

Subgroup analysis of the primary performance endpoint by center, and US vs OUS, will be used to evaluate the poolability of the results. The significance of center-to-center variability in treatment effect will be evaluated by including an interaction term of treatment group by center in a logistic regression model. In the case that poolability is questionable, the reasons for differential treatment effect, such as patient and clinical characteristics, will be investigated and reported.




#### 8 DATA MANAGEMENT

## 8.1 Data Capture

Data capture will be performed using an Electronic Data Collection (EDC) system in conjunction with electronic patient reported outcome collection tools implemented in the smartphone application. The clinical sites will use electronic case report forms (eCRFs) to document the information required by the study CIP.

The EDC provider is ClearClinica. The EDC allows for the secure collection, transmission, validation, monitoring and real-time administration of study data gathered at investigative sites, and by the patient via the smartphone application. The system allows password-restricted access to clinical trial information based on individuals' roles and responsibilities. The EDC is compliant with 21 CFR Part 11 and FDA's "Guidance: Computerized Systems Used in Clinical Trials."

Except for Patient Reported Outcome entered directly by the patient to the smartphone App, data reported on the eCRF should be driven from source documents and be consistent with these source documents. Editing of data is done under full audit trail.

PRO data collected from the smartphone applications will be saved in dedicated log files on the smartphones for backup purposes and transferred to the EDC system at end of study visit.

## 8.1.1 Direct Data Entry

For several CRF fields Source Data Verification (SDV) may not be possible as entries may not be found in source documents (e.g., migraine diary or other Patient Reported Outcome completed directly into the smartphone App). Therefore, it is allowed to use the CRF for direct data entry, but only for pre-defined fields.

## 8.2 Data Quality Assurance

To ensure the quality of clinical data across all subjects, a clinical data management review will be performed by sponsor on patient data submitted in the CRF. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the CIP and relevant regulations. To resolve any questions arising from the clinical data management review process, data queries and/or site notifications will be issued by sponsor. Discrepancy resolution will be documented within the database audit trail.

# 8.3 Electronic Signatures

The PI will electronically sign each individual eCRF after the data has been cleaned, monitored and data reviewed. The electronic signature asserts that the investigator inspected or reviewed the data on the eCRF, the data queries, and the site notifications, and agrees with the content. Any changes made to the data after electronic signature has been applied will result in invalidation of the original signature, and the PI will be required to re-sign the data after reviewing the change(s).



Protocol number: TCH-003


# 8.4 Verification, validation and securing of electronic data capture system

Verification and validation of the EDC and eCRFs will be performed by a team comprising representatives of the developer, the sponsor and at least one of the participating sites. Verification and validation report will be held by the sponsor.

#### 8.5 Records and Data Retention

Copy of all records (e.g., informed consent documents, source data, safety reports, study device dispensing records, etc.) which support case report forms for this study, will be retained in the files of the responsible investigator for a minimum of five (5) years following notification by the sponsor that all investigations (not merely the investigator's portion) are completed, terminated and/or discontinued. If the principal investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The sponsor must be notified in writing of the name and address of the new custodian within 5 days after such transfer occurs.

Database will be retained by the EDC system provider for a minimum of 5 years.

## 8.6 Other Aspects of Clinical Quality Assurance

Site PI or a person designated by the site PI is responsible for establishing and maintaining adherence to the study protocol. Study PI is responsible for addressing quality assurance issues (correcting procedures that are not in compliance with protocol). Study Coordinator is responsible for quality control issues (i.e. correcting errors in data entry).

Sponsor will assign a monitor to monitor the investigational sites throughout the study. All outstanding issues and findings that site personnel become aware of will be communicated and handled in agreement with Monitoring Plan.

Sponsor auditing of the site may be done before the completion of the study to ascertain data quality and integrity.

The Food and Drug Administration (FDA) and/or the local state health authorities may request access to all study records, including source documents, for inspection. The investigator and site staff agree to cooperate with these audits. The investigator must notify the sponsor of any health authority audit as soon as notification of such audit is made. A representative or designee of sponsor may be present during health authority audit.




#### 9 AMENDMENTS TO THE CLINICAL INVESTIGATION PLAN

The protocol is not to be amended by the investigator without first obtaining sponsor's approval. Amendments initiated by the sponsor, or initiated by the investigator and then approved by the sponsor, will be submitted for approval to local IRB/EC and, if applicable, to the respective Regulatory Authority (RA). Protocol amendments should receive the IRB/EC approval, and if submitted to the RA, a regulatory approval as well, prior to implementation in the study. For non-substantial changes (e.g. minor logistical or administrative changes, change of monitor(s), telephone numbers, renewal of insurance) not affecting the rights, safety and well-being of human subjects or not related to the clinical investigation objectives or endpoints, a simple notification to the IRB/EC and, where appropriate, regulatory authorities can be sufficient.

The following documents are relevant to the protocol, but are not considered part of the protocol. They are stored and modified separately. As such, modifications to these documents do not require protocol amendments.

- Site Roster
- Case report forms
- Data Management Plan
- Monitoring Plan
- Statistical Analysis Plan
- DMC



Protocol number: TCH-003


#### 10 CLINICAL INVESTIGATION PLAN DEVIATIONS

A protocol deviation is any noncompliance with the clinical study protocol, Good Clinical Practice, or related SOPs requirements. The noncompliance may be on the part of the subject, the investigator, or study staff.

The protocol is not to be deviated by the investigator or the co-investigators without first obtaining sponsor approval except in cases where the safety and well-being of a patient will be affected, as stated in section 4.5.4 b of the ISO 14155 (2011).

Compliance to the protocol will be assessed by study monitor during monitoring visits as well as remotely, using designated reports provided by the EDC system.

All deviations from the protocol will be addressed in study subject source documents and promptly reported to the site IRB, according to local requirements.

# 10.1 Procedures for Recording, Reporting and Analyzing Protocol Deviations

All protocol deviations need to be documented in source documents and appropriate eCRF.

The Study Monitor is responsible for identifying and reviewing protocol deviations with the investigator or designee and documenting the issue and action/outcome of the protocol deviation in the MVR and any follow up letter / communication to the principal investigator.

The Study Monitor will ensure that major protocol deviations are discussed with the Investigator. Major deviations are those deviations that:

- impact patient safety
- alter the risk/benefit ratio
- compromise the integrity of the study data
- affect willingness of the patient's participation in the study

Deviations will be reported to the IRB/EC periodically or as specified by local regulations. Further documentation of any changes in research activity should be submitted to the sponsor and the IRB/EC if:

- They are related to any instance of serious or continuing non-compliance with governing regulations/requirements of the IRB/EC, and/or
- Related to changes in protocol specified patient activity and procedures.

The Study Monitor will, in addition to the above immediate reporting, document all deviations in the monitoring visit report and follow-up letters. The monitor will discuss deviations with relevant site personnel. If needed, a Note to File will be issued and filed in the relevant file and a copy sent to sponsor.

Sponsor or its designee will review records of deviations and will consider the need for corrective and preventive action and further external reporting to regulatory authorities. Deviations will be




summarized and included in the study report. Assessment and discussion of their potential impact / lack of impact on study results will be addressed.

## 10.2 Notification Requirement and Timelines

Major deviations should be escalated to the sponsor within 5 business days.

Protocol deviations must be reported to local IRB/EC per their guidelines. The site PI or other designated site staff member is responsible for knowing and adhering to local IRB/EC requirements.




#### 11 DEVICE ACCOUNTABILITY

Devices will be provided by Theranica Bioelectronics (sponsor), bearing required labeling. Upon being handed to study participant, device number will be documented in CRF and in site log. Each batch of devices delivered to clinical sites for allocation to study participants is accompanied by a shipment note. Device shipment records are maintained by sponsor and on site.

Prior to distribution, the devices are stored in a designated locked cabinet. Access to investigational devices is controlled by the research staff. The devices are only used in the clinical investigation and according to the study protocol.

Each device has a sticker on it with a unique number. When a device is handed to a study participant, it is coupled to the participant's smartphone by means of Bluetooth connection.

In the course of device allocation, application installation and device – application connection establishment, site allocated User ID is entered by study coordinator via the Application.

The triplet of IDs (User ID, phone ID, device ID) provides means of identifying technical and PRO data from each participant in the electronic database while protecting participant's privacy.

The clinical investigator will be responsible for the safe storage of devices in accordance with instructions given by Theranica Bioelectronics, with restricted access to the investigational materials in their possession, thereby preventing use of any materials by any person not participating in the study. Device accountability records will be reviewed during monitoring visits.

The investigator will be responsible for providing device use training to the patients according to the IFU and protocol and for maintaining product inventory and records.

As part of study closure, all unused devices must be returned in their original packaging to Theranica Bioelectronics.




#### 12 STATEMENTS OF COMPLIANCE

This study will be conducted in compliance with the protocol (after being approved by the local EC and, if required, by the local RA), the Good Clinical Practice (GCP) per ISO 14155 (2011) standard and the ethical principles that have their origin in the Declaration of Helsinki.

The Informed Consent Form (ICF), patient's information material, and advertising material (if applicable) must be submitted and approved by the IRB/EC (and RA when needed), and any request by the IRB/EC or RA will be followed. Written approval of the protocol, ICF, patient's information material, and any advertising material (if applicable) must be obtained from the EC and if applicable the corresponding RA prior to any patient enrollment.

Adequate insurance policy will be held valid for the entire study duration as well as for the discovery period required per local regulation.




#### 13 INFORMED CONSENT PROCESS

Written informed consent must be obtained from each study patient prior to commencing any CIP-specific procedures. A written informed consent (approved by sponsor and the IRB/EC) must be signed and dated by the patient, and the person who conducted the informed consent discussion. Additionally, the person who conducted the informed consent discussion will indicate that Informed Consent has been obtained by noting so in the appropriate section of the. Patients will be given a copy of the signed informed consent document. The signed informed consent will be retained with the study records at the investigational site. New findings relevant to the patient's continued participation will be made available to the patients after approval of such updates by the IRB/EC.

Informed consent accurately describes all aspects of the clinical investigation that are relevant to the subject's decision to participate in the study.



Protocol number: TCH-003


#### 14 ADVERSE EVENTS

Capturing of adverse events will serve for safety evaluation.

Adverse events encountered during treatment will be captured via end of study questionnaire and interview.

This study will use the list in section 14.7 below for nomenclature of adverse events complications reported in the CRF for Device related side effects.

Non-Device adverse events will be graded according to section 14.2.1 below. AE resulting from a procedure that is not related to the device, are considered as general AEs.

On-site visits to investigate adverse events and follow them up will be scheduled at the discretion of the principal investigator. Unscheduled visits and termination visit will be reported using designated case report forms.

If at the last visit there will be a Device related AE/side effect that is still active, the patient will be followed to completion or until a steady state is achieved for a continuous period of 2 weeks.

.

## 14.1 Characteristics of an Adverse Event

#### 14.1.1 Severity of the Adverse Event

Severity of AEs will be determined using the following scale:

- Mild: The patient is aware of a sign or symptom, but it is easily tolerated
- Moderate: Discomfort or interference with usual activity
- Severe: Incapacitating, with inability to engage in usual activity

#### 14.1.2 Relationship of an AE and SAE to the Study Device

The relationship of the adverse event to the study device is defined as follows:

Definite: An adverse event has a definite determination that it was caused due to the device.

Probable: An adverse event has a strong temporal relationship to study device or recurs on rechallange, and another etiology is unlikely or significantly less likely.

Possible: An adverse event has a strong temporal relationship to study device, and an alternative etiology is equally or less likely compared to the potential relationship to study device.

Unrelated - The AE is clearly NOT related to the device.

# 14.2 Definitions of Adverse Event and Adverse Device Effect

An <u>adverse event (AE)</u> is any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in study participants, whether or not related to the investigational device. This should relate to baseline information whenever available.



Protocol number: TCH-003

Page **67** of **94** 

An adverse device effect (ADE) is an adverse event related to the use of the investigational device. In this study the ADE is refers to "side effect" or "complications".

## 14.3 Definition of Serious Adverse Event

A serious adverse event (SAE) is an adverse event, that

- a) led to death,
- b) led to serious deterioration in the health of the subject, that either resulted in
  - 1) a life-threatening illness or injury, or
  - 2) a permanent impairment of a body structure or a body function, or
  - 3) in-patient or prolonged hospitalization, or
  - 4) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
- c) led to fetal distress, fetal death or a congenital abnormality or birth defect

  It is responsibility of site PL to report any Serious Adverse Event or Serious Adverse

It is responsibility of site PI to report any Serious Adverse Event or Serious Adverse Device Event to the sponsor, within 24 hours to:

**Theranica Bioelectronics** 

Dr. Dagan Harris

Tel: +972.72.390.9758 Fax: + 972.72.390.9755

Email: dagah@theranica.com

A <u>Serious device related adverse effect</u> (SADE) is an adverse event related to the use of the investigational device and that is considered by regulations and definitions as Serious.

# 14.4 Device Deficiency

Device deficiency is an inadequacy with respect to the device's identity, quality, durability, reliability, safety, or performance, such as a malfunction, failure, use error or inadequate labeling. Device deficiencies may or may not be associated with an adverse event.

All device deficiencies will be entered in the eCRF. Device deficiencies that were associated with an SAE or that could have led to an SAE if a) suitable action had not been taken or b) intervention had not been made or c) if circumstance had been less fortunate, will be reported within 24 hours of occurrence. If possible, the device(s) associated with a malfunction or failure should be retained until arrangements for its collection are made by the sponsor.

Device deficiencies will be summarized and reported in the clinical study report and will be reported to the regulatory authorities per country's applicable reporting requirements.

# 14.5 Time-frame for Investigator Reporting AE to Sponsor, EC, RA

Serious adverse events, whether or not related to the device, and whether anticipated or unanticipated, must be reported to the sponsor within 24 hours of learning of the event occurrence by the site staff. This requirement is in addition to, and does not replace, other investigator responsibilities for adverse event reporting. Notification on a SAE is forwarded to




sponsor designated contact person. Additionally, SAEs should be reported by the site to the involved IRB/EC and Regulatory Authorities as applicable.

Unanticipated device related adverse events shall be reported to the sponsor within 48 hours of learning of the event occurrence by the site staff.

In addition, device related side effects shall be reported to the sponsor and documented in monitoring visit/phone call summary.

Any AE that results in withdrawal from observation in the study must be reported to the sponsor within 24 hours after the decision to withdraw the patient is made.

Any death occurring during the study must be reported to the sponsor within 24 hours of discovery of the event. "Death" should not be reported as an AE, the cause of death should be reported as an AE. The only exception is "Sudden Death" when the cause is unknown. A copy of the death records, death certificate and an autopsy report (if performed) must be provided to the sponsor as soon as possible.

The sponsor is responsible for relaying adequate information on SAEs to the regulatory authorities per country's applicable reporting requirements.

## 14.6 Adverse Event Reporting Forms

The eCRFs for AE or SAE will include all relevant information of the AE or SAE with regards to onset and resolution time, grade, causality to device, treatment given etc.

# 14.7 Foreseeable Complications and Anticipated Adverse Device Related Effects.

Possible adverse events associated with Transcutaneous Electrical Nerve Stimulation include, but are not limited to the following:

- Anxious mood
- Burn marks
- Increased air temperature sensitivity
- Itching
- Muscle fatigue
- Muscle spasms
- Skin irritation or redness
- Stinging sensations

The following migraine symptoms are foreseeable and will not be considered as device related: headache, nausea, light sensitivity, sensitivity to noise or odors, stomach upset, abdominal pain, loss of appetite, cold or heat sensation, paleness, fatigue, dizziness, fever (rare), blurred vision, vision symptoms such as bright flashing dots or lights, blind spots, wavy or jagged lines (aura).




## 14.8 Safety Monitoring and Adjudication of Adverse Events

The sponsor will review submitted AE information and may request supplemental information if needed. For SAE, USADE and ADE (as classified by the investigator) a narrative will be prepared and adjudicated for assessing the relatedness, seriousness and possible action items required. The sponsor may ask for further information or clarification from the investigator. A summary of the adjudication results will be issued; if different than investigator's report, PI will be notified.

Adjudicated events will serve as a basis for reporting AE/SAE. Differences between site-reported events and adjudicated events will also be presented and discussed in the report.




## 15 VULNERABLE POPULATION

No vulnerable population will be enrolled to this study.



Protocol number: TCH-003 

#### 16 EARLY TERMINATION OF THE CLINICAL INVESTIGATION

## 16.1 Criteria and Arrangements

The study may be discontinued if:

- At any time, in the opinion of study PI, the study represents an unreasonable medical risk to patients.
- The sponsor decides to terminate the study due to company considerations (e.g. Data Monitoring Committee recommends study termination based on futility analysis of interim data)

In the event of clinical investigation premature termination or suspension, sponsor will send a report outlining the circumstances to the corresponding IRB/EC, regulatory body and all investigators. A suspended or terminated clinical investigation may not be re-initiated without approval of the corresponding IRB/EC and relevant RA, as applicable. In the event of clinical investigation premature termination or suspension, enrolled subjects will be followed up as per the institution's standard of care.

## 16.2 Requirements for Patient Follow-Up in case of Withdrawal

In case of patient withdrawal, all efforts will be made to collect and report the final visit observations as thoroughly and timely as possible.



Protocol number: TCH-003 

## 17 PUBLICATION POLICY

The publication policy is defined in the sponsor – investigator agreement.



## 18 PATIENT CONFIDENTIALITY & DATA PROTECTION

The privacy of participants and confidentiality of personal data will be maintained in reports and publications and will not be otherwise published in any way.

Privacy will be maintained according to prevailing national data protection, privacy and secrecy laws. Each patient will be identified by a unique patient identification number.

However, the sponsor's monitor or representative and regulatory representatives, auditors and inspectors may have access to medical files in order to verify authenticity of data collected, as documented in informed consent form.




## 19 GUIDELINES AND APPLICABLE DOCUMENTS

- 1. EN ISO 14155; (2011): Clinical investigation of medical devices for human patients
- 2. EN ISO 14971; (2012): Medical devices Application of risk management to medical devices.



Protocol number: TCH-003 

#### 20 REFERENCES

1. Bloudek I. et al. Cost of healthcare for patients with migraine in five European countries: results from the International Burden of Migraine Study (IBMS). J Headache Pain (2012) 13:361–378

- Goadsby PJ, Lipton RB, Ferrari MD. Migraine current understanding and treatment. N Engl J Med, 346: 257
- 3. Martelletti et al. Neuromodulation of chronic headaches: position statement from the European Headache Federation. The Journal of Headache and Pain 2013, 14:86
- 4. Schoenen J et al., Migraine prevention with a supraorbital transcutaneous stimulator. Neurology 80 February 19, 2013
- 5. Magis D. et.al. Safety and patients' satisfaction of transcutaneous Supraorbital NeuroStimulation (tSNS) with the Cefaly® device in headache treatment: a survey of 2,313 headache sufferers in the general population. The Journal of Headache and Pain 2013, 14:95
- 6. Magis D, Schoenen PGJ, Transcutaneous Vagus Nerve Stimulation (tVNS) for headache prophylaxis: initial experience. The Journal of Headache and Pain 2013, 14(Suppl 1):198
- 7. Slavin KV, Nersesyan H, Wess C. Peripheral neurostimulation for treatment of intractable occipital neuralgia. Neurosurgery 2006; 58:112.
- 8. Ristić D, Ellrich J. Innocuous Peripheral Nerve Stimulation Shifts Stimulus—Response Function of Painful Laser Stimulation in Man. Neuromodulation 2014; 17: 686
- 9. Nir RR et.al. A psychophysical study of endogenous analgesia: the role of the conditioning pain in the induction and magnitude of conditioned pain modulation. Eur J Pain. 2011 May;15(5):491
- Burstein R, Cutrer MF, Yarnitsky D. The development of cutaneous allodynia during a migraine attack clinical evidence for the sequential recruitment of spinal and supraspinal nociceptive neurons in migraine. Brain. 2000 Aug;123 ( Pt 8):1703
- Lipton RB et. al. Single-pulse transcranial magnetic stimulation for acute treatment of migraine with aura: a randomized, double-blind, parallel-group, sham-controlled trial. The Lancet 2010; 9:373
- 12. Barbanti P et.al. Non-invasive vagus nerve stimulation for acute treatment of high-frequency and chronic migraine: an open-label study. The Journal of Headache and Pain. 2015 16:61
- 13. Machin, D., Campbell, M.J. Statistical Tables for Design of Clinical Trials Blackwell Scientific Publications, Oxford (1987)
- 14. Fleiss, J.L., Tytun, A., Ury, S.H.K. "A simple approximation for calculating sample sizes for




comparing independent proportions" Biometrics 36(1980) pp. 343-346

- 15. Allais G, De Lorenzo C, Quirico PE, Lupi G, Airola G, Mana O, Benedetto C. Non-pharmacological approaches to chronic headaches: transcutaneous electrical nerve stimulation, laser therapy and acupuncture in transformed migraine treatment. Neurol Sci. 2003 May; 24 Suppl 2: S138-42
- 16. Marchand S et.al. Is TENS purely a placebo effect? A controlled study on chronic low back pain Pain. 1993; 54(1):99-106.
- 17. Johnson MI, Ashton CH, Thompson JW. An in-depth study of long-term users of transcutaneous electrical nerve stimulation (TENS). Implications for clinical use of TENS. Pain. 1991; 44(3):221-9.
- 18. J.J. Amer-Cuenca. Programacio'n y aplicacio'n de la estimulacio'n nerviosa ele'ctrica transcuta'nea (TENS): gui'a de pra'ctica cli'nica basada en la evidencia. Fisioterapia 2010;32(6):271–278
- 19. Oosterhof J. Outcome of transcutaneous electrical nerve stimulation in chronic pain: short-term results of a double-blind, randomised, placebo-controlled trial. J Headache Pain (2006) 7:196–205
- 20. Chesterton LS et.al. Sensory stimulation (TENS): effects of parameter manipulation on mechanical pain thresholds in healthy human subjects. Pain 2002; 99:253-62.
- 21. Eton DT et. al. A systematic review of patient-reported measures of burden of treatment in three chronic diseases. Patient Related Outcome Measures 2013:4 7–20
- 22. Tran VT et. al. Adaptation and validation of the Treatment Burden Questionnaire (TBQ) in English using an internet platform. BMC Medicine 2014, 12:109
- 23. Lines CR, Vandormael K, Malbecq W. A comparison of visual analog scale and categorical ratings of headache pain in a randomized controlled clinical trial with migraine patients. Pain 93 (2001) 185±190
- 24. CR Mehta and SJ Pocock Adaptive Increase in Sample Size when Interim Results are Promising: A Practical Guide with Examples; Statistics in Medicine. 2000; 00:1–6
- 25. Chen et al., Increasing the sample size when the unblinded interim result is promising; Statistics in Medicine. 2004; 23:1023–1038
- 26. Broberg. Sample size re-assessment leading to a raised sample size does not inflate type I error rate under mild conditions; Medical Research Methodology 2013, 13:94
- 27. Younger J, McCue R., Mackey S.. Pain Outcomes: A Brief Review of Instruments and Techniques, Curr Pain Headache Rep. 2009 February; 13(1): 39–43



Protocol number: TCH-003


#### 21 ACRONYM LIST

ADE - Adverse Device Effect

AE - Adverse Event

CA – Competent Authority

CE - Conformité Européenne [CE Mark]

CI - Confidence Interval

CIP - Clinical Investigation Plan

CRF - Case Report Form

CV - Curriculum Vitae

d - Day

DM - Data Management

DNIC - diffused noxious inhibitory control

EC - Ethical Committee

GCP - Good Clinical Practice

**GMP- Good Manufacturing Practice** 

**IB** - Investigator Brochure

ICF - Informed Consent Form

ICH - International Conference on Harmonization

IFU - Instructions for Use

ISO - International Organization for Standardization

m - Month

MDD - Medical Device Directive

MoH - Ministry of Health

NPS - Numeric Pain Rating Scale

PI - Principal Investigator

PP - Per-Protocol analysis set

**PRO - Patient Reported Outcomes** 

RA - Regulatory Authority

SADE - Serious Adverse Device Effect

SAE - Serious Adverse Event




SD - Standard Deviation

SDV - Source Data Verification

**SOPs - Standard Operating Procedures** 

w - Week




# **APPENDIX A. STIMULATION PROGRAMS**

#### Active device:

• Modulated waveform:

• Biphasic, rectangular, symmetrical

• Pulse duration (μsec): 400

Pulse frequency (Hz): 100-120\*

• Max output current (mA): 60

 Modulating waveform: amplitude modulation at 2 Hz, with amplitude attenuation of 0.75.

#### Sham device:

• <u>Waveform:</u> rectangular, symmetrical

• Pulse duration (μsec): pseudo-random between 80 to 400

• Pulse frequency (Hz): 0.083 on average

• Max output current (mA): 40




# APPENDIX B. CASE REPORT FORMS LIST AND DRAFT CRF QUESTONS

Electronic CRFs are being implemented, so the tables below provide contents but not look of the planned forms.

The CRFs are comprised of the following forms:

| | eCRFs List |
|-----|----------------------------------|
| 1 | Demographics |
| 2 | Medical History |
| 3 | Migraine Assessment |
| 4 | Medical assessment |
| 5 | Eligibility (Incl./Excl.) |
| 5a | Informed consent |
| 6 | Device identification |
| 7 | Migraine Diary |
| 8 | Treatments and outcomes |
| 9 | Adverse Events |
| 9a | SAE |
| 10 | Protocol Deviations |
| 11 | Device deficiency |
| 12 | Concomitant Medication |
| 12a | Migraine Medication |
| 13 | End of Study Questionnaire |
| | Changes in medication during the |
| 13a | study period |
| 14 | Study exit form |

## 1. Demographics

| Question | Туре | Optional input | Part of eligibility criteria (Y/N) |
|---|---|---|---|
| Date of Birth | dd/mm/YYYY | | |
| Age at enrollment | | calculated | Υ |
| Gender | RadioButton | Male | |
| | | Female | |



| Protocol number: TCH-003 | Page <b>81</b> of <b>94</b> |
|--------------------------|-----------------------------|
|--------------------------|-----------------------------|

| Race (check one or | RadioButton | American Indian or Alaskan Native |
|---|---|---|
| specify other) | | Asian |
| | | African American |
| | | Native Hawaiian or other Pacific |
| | | Islander |
| | | Caucasian |
| | | African Arab |
| | | Eastern Arab |
| | | Other: |
| height | Open text<br>(number) | cm/inches( radio buttons) |
| weight | Open text<br>(number) | kg/pounds(radio buttons) |

## 2. Medical History

| Question | Туре | Optional input |
|---|---|---|
| Date of assessment | Date field | |
| Prior surgeries | Radio buttons | yes/no |
| If yes, year and reason | Open text | unknown |
| Other prior hospitalizations | Radio buttons | yes/no |
| If yes, year and reason | Open text | unknown |
| Which of the following conditions | Checkbox with multiple | Neurological |
| was the patient treated for in the | choices | Psychiatric |
| past? Check all that apply | | HEENT |
| | | Respiratory |
| | | Cardiovascular |
| | | Gastrointestinal/Hepatic |
| | | Renal |
| | | Genitourinary |
| | | Musculoskeletal |
| | | Dermatological |
| | | Hematological |
| | | Metabolic/Endocrine |
| | | Allergy |
| | | Other |
| If Other, please specify | Open text | |
| If any of the above checked, please | Open text | unknown |
| detail year diagnosed and specifics | | |
| Does the patient currently smoke or chew tobacco? | Radio buttons | yes/no |




| If yes, how many packs per day? | Open text (number) | |
|-------------------------------------|--------------------|--------|
| If no, had he/she in the past? | Radio buttons | yes/no |
| If yes, please specify year stopped | Open text | |
| If yes, please specify how many | Open text | |
| packs per day | | |
| Does the patient drinks alcohol, | Radio buttons | yes/no |
| beer or wine? | | |
| If yes, how many drinks per week? | Open text (number) | |
| If no, had he/she in the past? | Radio buttons | yes/no |
| If yes, please specify year stopped | Open text | |
| If yes, please specify how many | Open text | |
| drinks per week | | |

## 3. Migraine Assessment

| Question | Туре | Optional input | Part of eligibility criteria (Y/N) |
|---|---|---|---|
| Year of migraine diagnosis | drop down<br>list | unknown | |
| Average number of attacks per month | input field | | Υ |
| Average number of migraine days per month | input field | | Υ |
| Number of other types of headaches per month | radio buttons | "0" / "1-5" / "6 and<br>more" | |
| Use of preventive medication. If YES, fill in concomitant medication CRF entry | radio buttons | yes/no | |
| Any change in use/dose of preventive medication in the past two months | radio buttons | yes/no | Υ |
| How often do you experience aura preceding a migraine attack | radio buttons | Often /<br>Rarely /<br>None | |
| Average attack duration w/o medication | dropdown list | 0-2/ 2-6/ 6-12/ 12-<br>24/ 24-48/ More<br>than 48 | |




| Maximum pain level for an average attack, without medication (pain grade) | radio buttons | mild/moderate/se<br>vere | |
|---|---|---|---|
| Use of acute medication to treat the headache during migraine attack | dropdown list | always/sometime<br>s/rarely/never | |
| If yes, medication name | dropdown list | see rescue<br>medication list<br>sheet | |
| If yes, medication dose | fractional number | 23.5 | |
| If yes, medication dose units | radio buttons | mg/cc/other | |
| "if other, specify" - an input text window | input field | | |
| How long after pain start is rescue medication taken, on average | dropdown list | 0-20min/20-<br>40min, 40-<br>60min/1-2h/2-<br>4h/more than 4h | |
| Average attack duration with rescue medication | dropdown list | 0-2/ 2-6/ 6-12/ 12-<br>24/ 24-48/ More<br>than 48 | |
| Typical pain level for an average attack, 2 hours after rescue medication taken | None (0)<br>Mild (1)<br>Moderate (2)<br>Severe (3) | pain grade | |
| Migraine pain side | radio buttons | left/right/alternatin<br>g/both | Υ |
| Nausea/vomiting during attack | radio buttons | yes/no/sometime<br>s | Υ |
| Light sensitivity during attack | radio buttons | yes/no/sometime<br>s | Υ |
| Sound sensitivity during attack | radio buttons | yes/no/sometime<br>s | Υ |
| Where does your skin become more sensitive to touch or pressure when you have migraine | checkboxes | None<br>Scalp<br>Eye and/or<br>forehead<br>Body | Υ |




| | | nausea/light/nois |
|--------------------------|---------------|-------------------|
| Most bothersome migraine | | e/skin |
| symptom beyond pain | dropdown list | sensitivity/none |

#### 4. Medical assessment

| Question | Туре | Optional input | Part of eligibility criteria (Y/N) |
|---|---|---|---|
| Open wounds or burns, or irritated skin on upper arm area | Radio buttons | yes/no | n |
| Pregnancy test taken | Radio<br>buttons | yes/no/NA | |
| if no, specify reason | open text | | |
| Pregnancy test result | Radio buttons | positive/negative | |
| General motor and sensory function | Radio buttons | normal/abnormal | |

5. Eligibility

| Question | Туре | Optional input |
|---|---|---|
| Inclusion criteria | | |
| If any inclusion criterion is checked <b>No</b> , the patient i cannot be enrolled. | s considered ineligil | ole for this study and |
| Subject is 18-75 years old | Radio buttons | yes/no |
| Meets the ICHD-3 diagnostic criteria for migraine with and without aura | Radio buttons | yes/no |
| Subjects report 2-8 migraine attacks per month | Radio buttons | yes/no |
| Stable migraine preventive medications in the last two months prior to recruitment (No change in usage or dosage). | Radio buttons | yes/no |
| Subjects must be able and willing to comply with the protocol | Radio buttons | yes/no |
| Subjects must be able and willing to provide written informed consent protocol | Radio buttons | yes/no |
| Exclusion criteria | | |
| If any Exclusion criterion is checked <b>Yes,</b> the patient cannot be enrolled. | is considered inelig | ible for this study an |




| Subject has other significant pain, medical or psychologic problems that in the opinion of the | Radio buttons | yes/no |
|---|---|---|
| investigator may confound the study assessments | | |
| Subject has an implanted electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagus nerve neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator cochlear implant, Sphenopalatine | Radio buttons | yes/no |
| ganglion stimulator or Occipital nerve stimulator). | | |
| Subject has known uncontrolled epilepsy. | Radio buttons | yes/no |
| Any use of Cannabis including medical use. | Radio buttons | yes/no |
| Subject has >10 headache days per month. | Radio buttons | yes/no |
| Subject has undergone nerve block (occipital or | Radio buttons | yes/no |
| other) in the head or neck within the last 2 weeks. | Radio buttons | yes/no |
| Subject is participating in any other clinical study. | Radio buttons | yes/no |
| The subject does not have the basic cognitive and motor skills needed to operate a smartphone. | Radio buttons | yes/no |
| Pregnant, or trying to get pregnant | Radio buttons | yes/no/NA |
| Subject is experiencing a menstrually related migraine | Radio buttons | yes/no/NA |
| Received OnabotulinumtoxinA or any botulinum toxin injections for migraine within the previous month | Radio buttons | yes/no |
| Received parenteral infusions for migraine within the previous 2 weeks. | Radio buttons | yes/no |
| Subject participated in a previous study with the Nerivio Migra 1 device | Radio buttons | yes/no |
| Is patient eligible for participating in the study? ( If NO, patient should not be enrolled) | Radio buttons | Yes/No |

## 5a. Informed Consent

| Question | Туре | Optional input |
|---|---|---|
| Has the patient received written and oral explanation of the study? | Radio buttons | Yes/No |
| ICF version : | integer | number 1-10 |
| Date obtained and signed | dd/mm/YYYY | |




| Has the patient received a copy of the signed ICF? | Radio buttons | Yes/No |
|----------------------------------------------------|---------------|--------|
| If NO, explain why | Open text | |

## 6. Device identification

| Question | Туре | Optional input |
|---------------------|---------------|-------------------------------------|
| Smartphone ID | | fed from 1st connect event with app |
| Phone_ype | | fed from 1st connect event with app |
| Application Version | | fed from 1st connect event with app |
| SEW5120Ver | | fed from 1st connect event with app |
| Training - diary | radio buttons | fed from server when executed |

## 7. Migraine Diary

| | For each reported attack | | | |
|---|---|---|---|---|
| Attack<br>start | Attack number | sequential<br>number of this<br>attack in diary list | from server | |
| | Date and time | | from server | |
| | time elapsed after previous reported attack | dd/hh/mm | from server | dd/hh/mm |
| | Current migraine pain level | Current migraine pain level in pain grade categories | Radio buttons | Mild (1), Moderate (2),<br>Severe (3). |
| | Time from onset of | Time from onset | Dropdown list | under 30 minutes |
| | migraine pain | of migraine pain | | 30-60 minutes |
| | | | | over 60 minutes |
| | Nausea | Presence of nausea | Radio buttons | yes/no |
| | Sensitivity to light | Presence of photophobia | Radio buttons | yes/no |
| | Sensitivity to sound | Presence of phonophobia | Radio buttons | yes/no |
| | Increased skin sensation | Presence of allodynia | Radio buttons | yes/no |
| | MBS | most boresome symptoms | Radio buttons | Nausea/Photophobia/Pho<br>nophobia/Allodynia/None |
| | aura | | Radio buttons | yes/no |




| Status at 2h | Date and time | date and time | | |
|---|---|---|---|---|
| at Zn | | when record received | | |
| | Attack number | sequential<br>number of this<br>attack in diary list | from server | |
| | Migraine pain level 2 hours past attack start | Current migraine pain level in pain grade categories | Dropdown list | No pain (0), Mild (1),<br>Moderate (2), Severe (3). |
| | Medication | Whether rescue<br>medication was<br>taken | Radio buttons | yes/no |
| | Rescue medication name | Rescue<br>medication name | Free text from App | See Appendix 5.3 |
| | if medication has | | Radio buttons | Before start of treatment |
| | being used | | | Less than 2 hours after start of treatment 2 hours or more from |
| | | | | starting the treatment |
| | Nausea | Presence of nausea | Radio buttons | yes/no |
| | Sensitivity to light | Presence of photophobia | Radio buttons | yes/no |
| | Sensitivity to sound | Presence of phonophobia | Radio buttons | yes/no |
| | Increased skin sensation | Presence of allodynia | Radio buttons | yes/no |
| Status<br>at 48h | Attack number | sequential<br>number of this<br>attack in diary list | from server | |
| | Date and time | date and time<br>when record<br>received | from server | |
| | Migraine pain level<br>48 hours past attack<br>start | Current migraine pain level in pain grade categories | Dropdown list | No pain (0), Mild (1),<br>Moderate (2), Severe (3). |
| | Additional medication taken (after reported @2h) | Whether rescue<br>medication was<br>taken | Radio buttons | yes/no |
| | Rescue medication name | Rescue<br>medication name | Free text from App | See Appendix 5.3 |

#### 8. Randomization




| Question | Туре | Optional input |
|----------------------|---------------|-------------------------------------|
| Device ID | | fed from 1st connect event with app |
| Smartphone ID | | fed from 1st connect event with app |
| Phone_type | | fed from 1st connect event with app |
| Application_Version | | fed from 1st connect event with app |
| SEW5120Ver | | fed from 1st connect event with app |
| Training - treatment | radio buttons | fed from server when executed |

## 9. Treatment

| | Item | Description | Control type<br>for PRO | Values range |
|---|---|---|---|---|
| | Attack number | sequential number of<br>this attack in treated<br>attacks list | from server | |
| Attack | Date and time | | from server | |
| start | time elapsed after<br>previous reported<br>attack | dd/hh/mm | from server | dd/hh/mm |
| | Current migraine pain level | Current migraine pain level in pain grade categories | Radio<br>buttons | Mild (1), Moderate (2),<br>Severe (3). |
| | Time from onset of | Time from onset of | Dropdown | under 30 minutes |
| | migraine pain | migraine pain | list | 30-60 minutes |
| | | | | over 60 minutes |
| | Nausea | Presence of nausea | Radio<br>buttons | yes/no |
| | Sensitivity to light | Presence of photophobia | Radio<br>buttons | yes/no |
| | Sensitivity to sound | Presence of phonophobia | Radio<br>buttons | yes/no |
| | Increased skin sensation | Presence of allodynia | Radio<br>buttons | yes/no |
| | Aura | Presence of aura | Radio<br>buttons | yes/no |
| Status at<br>2h | Date and time | date and time when record received | | |
| | Attack number | sequential number of<br>this attack in treated<br>attacks list | from server | |




| | Current migraine pain level | Current migraine pain level in pain grade categories | Dropdown<br>list | No pain (0), Mild (1),<br>Moderate (2), Severe<br>(3). |
|---|---|---|---|---|
| | Medication | Whether rescue<br>medication was<br>taken | Free Text | Yes/No |
| | Rescue medication name | Rescue medication name | Dropdown<br>list | See Appendix 5.3 |
| | if medication has being used | | Radio<br>buttons | Before start of treatment |
| | | | | Less than 2 hours after start of treatment |
| | | | | 2 hours or more from starting the treatment |
| | Nausea | Presence of nausea | Radio<br>buttons | yes/no |
| | Sensitivity to light | Presence of photophobia | Radio<br>buttons | yes/no |
| | Sensitivity to sound | Presence of phonophobia | Radio<br>buttons | yes/no |
| | Increased skin sensation | Presence of allodynia | Radio<br>buttons | yes/no |
| | MBS | most boresome symptoms | Radio<br>buttons | Nausea/Photophobia/P<br>honophobia/Allodynia/<br>None |
| Status at<br>48h | Date and time | date and time when record received | | |
| | Attack number | sequential number of<br>this attack in treated<br>attacks list | from server | |
| | Current migraine pain level | Current migraine pain level in pain grade categories | Dropdown<br>list | No pain (0), Mild (1), Moderate (2), Severe (3). |
| | Additional medication taken (after reported @2h) | Whether rescue<br>medication was<br>taken | Radio<br>buttons | yes/no |
| | Rescue medication name | Rescue medication name | Free Text | See Appendix 5.3 |

## 10. Treatment summary

| Item | Description | Control | type | Values range |
|------|-------------|---------|------|--------------|
| | | for PRO | | |



| qualified | Radio buttons | yes/no |
|---|---|---|
| treatment status | Radio buttons | completed/aborted/stopped/unknown |
| report status | Radio buttons | missing data/evaluable/complete |
| average<br>stimulation<br>intensity | from server | |
| max stimulation intensity | from server | |
| treatment<br>duration | from server | |

#### 11. Phone call

| Question | Туре | Optional input |
|---|---|---|
| Date | Date field | |
| Time | time filed | |
| Alert performed for ? | Radio buttons | mising 2 hours feedback missing 48 hours feedback Battery level below 40% Battery level below 25% Battery level below 10% Low stimulation intensity level Repeated abort or incompletion of the qualified session Long inactive/off-line time Less than 2 qualified attacks per month |
| Subject contacted? | Radio buttons | Yes/No |
| Call effective? | Radio buttons | Yes/No |
| Comments | Open text | |

# 12. End of Study questionnaire

| Question | Туре | Optional input |
|---|---|---|
| Usability assessment: How easy was it to administer treatment | Dropdown<br>list | very easy (1), easy (2), neutral (3), uncomfortable (4), difficult (5) |
| Blinding assessment: which group do you think you were assigned? | Dropdown<br>list | active/sham/do not know |
| Global impression of change: please rate your current status | Dropdown<br>list | very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse |




| | (5), much worse (6), or (7) very much worse |
|-------|---------------------------------------------|
| Radio | yes/no |
| | Radio<br>buttons |

#### 13. Study exit form

| Question | Туре | Optional input |
|---|---|---|
| Date of study termination | Date field | |
| Did the patient complete the | Radio buttons | yes |
| study according to the protocol ? | | no |
| If no, select from the list: | Dropdown list | Roll in screen failure |
| | | Patient withdrew consent |
| | | Adverse event or SAE |
| | | Noncompliance with the protocol |
| | | Lost to follow up |
| | | Other |
| If other, please specify | Open text | |
| Subject received | Radio buttons | Yes/No |
| compensation | | |
| Additional comments | Open text | |
| log files copied | Radio buttons | Yes/No |

## 14. Concomitant medications

| PRIMARY QUESTION | | |
|---|---|---|
| Is the subject taking any medication that will be continued during the study? | Radio buttons | yes/no |
| GRID | | |
| Question | Туре | Optional input |
| Migraine related? | Radio buttons | yes/no |
| Medication name | Open text | |
| If Related to migraine, Use ? | Radio buttons | preventive/rescue |
| If Not Related to migraine, Administered for | Open text | |



| Protocol number: TCH-003 | Page <b>92</b> of <b>94</b> |
|--------------------------|-----------------------------|
|--------------------------|-----------------------------|

| If Related to AE/ SAE then AE/ SAE Number: | Open text | |
|---|---|---|
| | (number) | |
| Daily dose | fractional number | 23.5 |
| Units | Radio buttons | cc, mg, other |
| if other unit, specify: | Open text | |
| Start date | Date field | |
| Stop/End date | Date field | |
| on going/unknown | Checkbox | |

#### 15. AE

| 15. AE | | |
|---|---|---|
| adverse event seq number | Open text | |
| Date of adverse event | Date field | |
| Date of report | Date field | |
| Initial or follow-up data | Radio | Initial report |
| | buttons | Follow-up data |
| Diagnosis | Open text | |
| Description | Open text | |
| Severity | Radio | Mild |
| | buttons | Moderate |
| | | Severe |
| Worsened pre-existing condition | Radio | Yes |
| | buttons | No |
| Relationship to study device | Dropdown | Not related |
| | list | Possibly related |
| | | Probably related |
| | | Definitely related |
| Relation to other therapy | Radio | Not related |
| | buttons | Possibly related |
| | | Probably related |
| | | Definitely related |
| If related to other therapy, please explain in the description above | Open text | |
| Action taken | Checkbox | None |
| | | Medication |
| | | Intervention |
| | | device treatment |
| | | discontinuation |
| | | Other |
| If intervention, please specify | Open text | |



Protocol number: TCH-003 

| If Other, please specify | Open text | |
|---------------------------------|------------|------------------------|
| Outcome | Radio | Resolved |
| | buttons | Resolved with sequelae |
| | | Ongoing, improved |
| | | Ongoing, unchanged |
| | | worsening |
| If resolved, date | Date field | |
| If resolved with sequelae, date | Date field | |
| Upload supporting information | Upload | |
| | file | |
| Study discontinued ? | Radio | Yes |
| | buttons | No |

## 16. SAE

| Item | Description | Values range |
|---|---|---|
| SAE number | Open text | |
| Date of adverse event | Date field | |
| End date | Date field | ongoing |
| Date of report | Date field | |
| Initial or follow-up data | Radio buttons | Initial report |
| | | Follow-up data |
| Diagnosis | Open text | |
| Description | Open text | |
| Severity | Radio buttons | Mild |
| | | Moderate |
| | | Severe |
| Was the adverse event serious | Radio buttons | Yes |
| (SAE)? | | No |
| If serious, specify | Radio buttons | Fatal |
| | | Immediately life |
| | | threatening |
| | | Required hospitalization or prolonged hospitalization |
| | | Persistent or significant disability/incapacity |
| | | Congenital anomaly/birth |
| | | defect |
| | | Other medically important |
| | | serious event |



Protocol number: TCH-003 

| If selected hospitalized: | date of hospitalization | Date field |
|---|---|---|
| | date of discharge | Date field |
| If selected Other medically important serious event, Specify: | Open text | |
| Worsened pre-existing condition | Radio buttons | Yes |
| | | No |
| Relationship to study device | Radio buttons | Not related |
| | | Possibly related |
| | | Probably related |
| | | Definitely related |
| Relation to other therapy | Radio buttons | Not related |
| | | Possibly related |
| | | Probably related |
| | | Definitely related |
| If related to other therapy, please explain in the description above | | |
| Action taken | Radio buttons | None |
| | | Medication |
| | | Hospitalization |
| | | Intervention |
| | | Other |
| If intervention, please specify | Open text | |
| If Other, please specify | Open text | |
| Outcome | Checkbox | Resolved |
| | | Resolved with sequelae |
| | | Ongoing, improved |
| | | Ongoing, unchanged |
| | | worsening |
| | | Fatal |
| If death, date | Date field | |
| If resolved, date | Date field | |
| If resolved with sequelae, date | Date field | |
| Upload supportive information | Upload file | |